CLINICAL TRIAL: NCT02719574
Title: A Phase 1/2, Multicenter, Open-label Study of FT-2102 as a Single Agent and in Combination With Azacitidine or Cytarabine in Patients With Acute Myeloid Leukemia or Myelodysplastic Syndrome With an IDH1 Mutation
Brief Title: Open-label Study of FT-2102 With or Without Azacitidine or Cytarabine in Patients With AML or MDS With an IDH1 Mutation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Forma Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2102-HEM-101
Record Dates: First submitted 2016-03-21; First posted 2016-03-25 (Estimated); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Acute Myeloid Leukemia; Acute Myelogenous Leukemia; Myelodysplastic Syndrome
Keywords: AML; MDS; IDH1; IDH
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — olutasidenib; Azacitidine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (11):
- PH1 Dose Escalation & Expansion FT-2102 (olutasidenib) (Experimental)
  Interventions: Drug: FT-2102 (olutasidenib)
- PH1 Esc. and Exp. FT-2102 (olutasidenib)+Azacitidine (Experimental)
  Interventions: Drug: FT-2102 (olutasidenib); Drug: Azacitidine
- PH1 Esc. and Exp. FT-2102 (olutasidenib)+Cytarabine (Experimental)
  Interventions: Drug: FT-2102 (olutasidenib); Drug: Cytarabine
- PH2 Cohort 1 FT-2102 (olutasidenib) Single Agent (Experimental): Relapsed or Refractory (R/R) AML
  Interventions: Drug: FT-2102 (olutasidenib)
- PH2 Cohort 2 FT-2102 (olutasidenib) Single Agent (Experimental): AML in morphologic complete remission or complete remission with incomplete blood count recovery (CR/CRi) after prior therapy with residual IDH1-R132 mutation
  Interventions: Drug: FT-2102 (olutasidenib)
- PH2 Cohort 3 FT-2102 (olutasidenib) Single Agent (Experimental): R/R AML/MDS, previously treated with FT-2102
  Interventions: Drug: FT-2102 (olutasidenib)
- PH2 Cohort 4 FT-2102 (olutasidenib)+Azacitidine (Experimental): R/R AML/MDS that are naïve to prior hypomethylating therapy and IDH1 inhibitor therapy
  Interventions: Drug: FT-2102 (olutasidenib); Drug: Azacitidine
- PH2 Cohort 5 FT-2102 (olutasidenib)+Azacitidine (Experimental): R/R AML/MDS that have inadequately responded to or have progressed on prior hypomethylating therapy
  Interventions: Drug: FT-2102 (olutasidenib); Drug: Azacitidine
- PH2 Cohort 6 FT-2102 (olutasidenib)+Azacitidine (Experimental): R/R AML/MDS that have been previously treated with single-agent FT-2102 as their last therapy prior to study enrollment
  Interventions: Drug: FT-2102 (olutasidenib); Drug: Azacitidine
- PH2 Cohort 7 FT-2102 (olutasidenib) Single Agent (Experimental): Treatment naïve AML for whom standard treatments are contraindicated
  Interventions: Drug: FT-2102 (olutasidenib)
- PH2 Cohort 8 FT-2102 (olutasidenib)+Azacitidine (Experimental): Treatment naïve AML who are candidates for azacitidine first line treatment
  Interventions: Drug: FT-2102 (olutasidenib); Drug: Azacitidine

INTERVENTIONS:
Drug: FT-2102 (olutasidenib) — FT-2102 (olutasidenib) will be supplied as 50 mg or 150 mg capsules and will be administered per the protocol defined frequency and dose level
Drug: Azacitidine — azacitidine will be administered per site's standard of care
  Other Names: Vidaza
  Arms: PH1 Esc. and Exp. FT-2102 (olutasidenib)+Azacitidine; PH2 Cohort 4 FT-2102 (olutasidenib)+Azacitidine; PH2 Cohort 5 FT-2102 (olutasidenib)+Azacitidine; PH2 Cohort 6 FT-2102 (olutasidenib)+Azacitidine; PH2 Cohort 8 FT-2102 (olutasidenib)+Azacitidine
Drug: Cytarabine — low-dose cytarabine will be administered per site's standard of care
  Arms: PH1 Esc. and Exp. FT-2102 (olutasidenib)+Cytarabine

SUMMARY:
This Phase 1/2 study will evaluate the safety, efficacy, PK, and PD of FT-2102 (olutasidenib) as a single agent or in combination with azacitidine or cytarabine. The Phase 1 stage of the study is split into 2 distinct parts: a dose escalation part, which will utilize an open-label design of FT-2102 (olutasidenib) (single agent) and FT-2102 (olutasidenib) + azacitidine (combination agent) administered via one or more intermittent dosing schedules followed by a dose expansion part. The dose expansion part will enroll patients in up to 5 expansion cohorts, exploring single-agent FT-2102 (olutasidenib) activity as well as combination activity with azacitidine or cytarabine. Following the completion of the relevant Phase 1 cohorts, Phase 2 will begin enrollment. Patients will be enrolled across 8 different cohorts, examining the effect of FT-2102 (olutasidenib) (as a single agent) and FT-2102 (olutasidenib) + azacitidine (combination) on various AML/MDS disease states.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven acute myeloid leukemia (AML) (except acute promyelocytic leukemia [APL] with the t(15;17) translocation) or intermediate, high-risk, or very high risk Myelodysplastic Syndrome (MDS) as defined by the World Health Organization (WHO) criteria or Revised International Prognostic Scoring System (IPSS-R) which is relapsed or refractory (R/R) to standard therapy and/or for which standard therapy is contraindicated or which has not adequately responded to standard therapy.
* Patients must have documented IDH1-R132 gene-mutated disease as evaluated by the site
* Good performance status
* Good kidney and liver function

Exclusion Criteria:

* Patients with symptomatic central nervous system (CNS) metastases or other tumor location (such as spinal cord compression, other compressive mass, uncontrolled painful lesion, bone fracture, etc.) necessitating an urgent therapeutic intervention, palliative care, surgery or radiation therapy
* Congestive heart failure (New York Heart Association Class III or IV) or unstable angina pectoris. Previous history of myocardial infarction within 1 year prior to study entry, uncontrolled hypertension or uncontrolled arrhythmias
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2016-04-30 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2024-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (60):
- United States (19):
  - UCLA Medical Center, Los Angeles, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Yale University, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York Medical College, Hawthorne, New York
  - Columbia University Medical Center, New York, New York
  - Cornell University Weill Medical College, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Sarah Cannon Research Institute - Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
- Australia (5):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Victoria Cancer Care Center, Parkville, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Box Hill Hospital, Monash University and Eastern Health Clinical School, Box Hill
- Princess Margaret Hospital, Toronto, Ontario, Canada
- France (11):
  - Service d'Hématologie Clinique, Hôpital Avicenne-APHP-Université Paris, Bobigny
  - Assistance Publique Hopitaux de Marseille (AP-HM) - Hopital Nord, Marseille
  - Centre Hospitalier Universitaire Nantes, Nantes
  - Hôpital Saint-Louis, Paris
  - Hopitaux Universitaires Est Parisien Hopital Saint-Antoine, Paris
  - Centre Hospitalier Universitaire (CHU) Bordeaux - Hospitaux du Haut Leveque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - University Hospital of Rennes, Rennes
  - Institut Universitaire du Cancer Toulouse - Oncopole, Toulouse
  - Centre Hospitalier Universitaire de Nancy - Hopital Brabois, Vandœuvre-lès-Nancy
  - Institut de Cancérologie Gustave Roussy, Villejuif
- Germany (4):
  - Staedtisches Klinikum Braunschweig gGmbH, Braunschweig
  - Universitaetsklinikum Giessen und Marburg GmbH - Klinik fuer Innere Medizin, Giessen
  - Landeszentrum fuer Zell- und Gentherapie, Halle
  - Universitätsklinikum Münster Medizinische Klinik A, Hämatologie, Hämostaseologi, Münster
- Italy (7):
  - AOU S. Luigi Gonzaga - Orbassano, Orbassano, Turin
  - Ospedale Mazzoni - UOC Ematologia Ascoli Piceno, Ascoli Piceno
  - Universita di Bologna, Bologna
  - Dipartimento di Oncologia Medica - IRST IRCC, Meldola
  - Università degli Studi di Parma, Parma
  - U.O. Ematologia Ravenna, Ravenna
  - Hospital Rimini Hematology, Department of Oncology and Hematoloy, Rimini
- South Korea (2):
  - Seoul National University Bundang Hospital, Gumi
  - Seoul National University Hospital, Seoul
- Spain (6):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Institut Català d'Oncologia-Hospital Duran i Reynals, Barcelona
  - Hospital Universitario 12 De Octubre, Madrid
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital La Fe, Valencia
- United Kingdom (5):
  - University College London Hospitals NHS Foundation Trust, London
  - St. George's University Hospital, London
  - Churchill Hospital, Oxford
  - Southampton General Hospital, Southampton
  - Royal Marsden Hospital, Sutton

REFERENCES:
- [Derived] Cortes J, Curti A, Fenaux P, Jonas BA, Krauter J, Montesinos P, Recher C, Taussig DC, Wang ES, Watts J, Wei A, Yee KW, Tian H, Sheppard A, Marzac C, de Botton S. Olutasidenib for mutated IDH1 acute myeloid leukemia: final five-year results from the phase 2 pivotal cohort. J Hematol Oncol. 2025 Nov 14;18(1):102. doi: 10.1186/s13045-025-01751-w. PMID 41239466
- [Derived] Cortes JE, Yang J, Roboz GJ, Dinner SN, Wang ES, Wei AH, Tian H, di Trapani F, Baer MR, Donnellan W, Watts JM. Olutasidenib alone or combined with azacitidine in patients with mutant IDH1 myelodysplastic syndrome. Blood Adv. 2025 Oct 28;9(20):5293-5305. doi: 10.1182/bloodadvances.2025016718. PMID 40668616
- [Derived] Cortes JE, Roboz GJ, Baer MR, Jonas BA, Schiller GJ, Yee K, Ferrell PB, Yang J, Wang ES, Blum WG, Mims A, Tian H, Sheppard A, de Botton S, Montesinos P, Curti A, Watts JM; Olutasidenib Combination Therapy Study Group. Olutasidenib in combination with azacitidine induces durable complete remissions in patients with relapsed or refractory mIDH1 acute myeloid leukemia: a multicohort open-label phase 1/2 trial. J Hematol Oncol. 2025 Jan 16;18(1):7. doi: 10.1186/s13045-024-01657-z. PMID 39819505
- [Derived] de Botton S, Fenaux P, Yee K, Recher C, Wei AH, Montesinos P, Taussig DC, Pigneux A, Braun T, Curti A, Grove C, Jonas BA, Khwaja A, Legrand O, Peterlin P, Arnan M, Blum W, Cilloni D, Hiwase DK, Jurcic JG, Krauter J, Thomas X, Watts JM, Yang J, Polyanskaya O, Brevard J, Sweeney J, Barrett E, Cortes J. Olutasidenib (FT-2102) induces durable complete remissions in patients with relapsed or refractory IDH1-mutated AML. Blood Adv. 2023 Jul 11;7(13):3117-3127. doi: 10.1182/bloodadvances.2022009411. PMID 36724515
- [Derived] Watts JM, Baer MR, Yang J, Prebet T, Lee S, Schiller GJ, Dinner SN, Pigneux A, Montesinos P, Wang ES, Seiter KP, Wei AH, De Botton S, Arnan M, Donnellan W, Schwarer AP, Recher C, Jonas BA, Ferrell PB Jr, Marzac C, Kelly P, Sweeney J, Forsyth S, Guichard SM, Brevard J, Henrick P, Mohamed H, Cortes JE. Olutasidenib alone or with azacitidine in IDH1-mutated acute myeloid leukaemia and myelodysplastic syndrome: phase 1 results of a phase 1/2 trial. Lancet Haematol. 2023 Jan;10(1):e46-e58. doi: 10.1016/S2352-3026(22)00292-7. Epub 2022 Nov 10. PMID 36370742

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total 336 participants enrolled in the study. In phase I, 78 participants were enrolled in single cohorts (FT-2102) and combination cohorts (FT-2102 with azacitidine/cytarabine) and in phase 2, 258 participants were enrolled in single cohorts (FT-2102) and combination cohorts (FT-2102 with azacitidine).
Pre-assignment Details: This study is comprised of 3 stages: A Phase 1 dose-escalation stage, a Phase 1 dose-expansion stage, and a Phase 2 stage. Participants with relapsed or refractory (R/R) acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS) with IDH1-R132 mutations received olutasidenib (FT-2102) alone or with azacitidine/ cytarabine in Phase 1 and 2. Based on the totality of data from Phase 1, Recommended Phase 2 dose (RP2D) for single-agent and combination treatment was determined.
Groups:
- Phase 1: FT-2102 100mg QD (Single Agent; Dose Escalation): Participants with AML or MDS received single agent of FT-2102 100 milligram (mg) orally once daily (QD) in 28-day cycles until MTD or MED achieved.
- Phase 1: FT-2102 150mg QD (Single Agent; Dose Escalation): Participants with AML or MDS received single agent of FT-2102 150 mg orally QD in 28-day cycles until MTD or MED achieved.
- Phase 1: FT-2102 150mg BID (Single Agent; Dose Escalation); Phase 1: FT-2102 150mg BID (Single Agent; Dose Expansion): Participants with AML or MDS received single agent of FT-2102 150 mg orally BID in 28-day cycles until MTD or MED achieved.
- Phase 1: FT-2102 300mg QD (Single Agent; Dose Escalation): Participants with AML or MDS received single agent of FT-2102 300 mg orally QD in 28-day cycles until MTD or MED achieved.
- Phase 1: FT-2102 150mg QD+Azacitidine (Combination Therapy; Dose Escalation): Participants with AML or MDS received combination therapy (FT-2102 150 mg QD and azacitidine administered at the dose of 75 mg/m^2 for 7 days IV/SC per every 28-day cycle) until treatment discontinuation.
- Phase 1: FT-2102 150mg BID+Azacitidine (Combination Therapy; Dose Escalation); Phase 1: FT-2102 150mg BID+Azacitidine (Combination Therapy; Dose Expansion): Participants with AML or MDS received combination therapy (FT-2102 150 mg BID and azacitidine administered at the dose of 75 mg/m^2 for 7 days IV/SC per every 28-day cycle) until treatment discontinuation.
- Phase 1: FT-2102 150mg BID+ Cytarabine (Combination Therapy; Dose Expansion): Participants with AML harboring IDH1 mutation received FT-2102 150 mg BID in combination with low-dose cytarabine (LDAC) administered at the dose of 20 mg BID SC for 10 days every 28-day cycle until treatment discontinuation.
- Phase 2: Cohort 1; FT-2102 (Single Agent): Participants with relapsed/refractory (R/R) AML received single agent of FT-2102 150 mg BID in continuous 28-day cycles.
- Phase 2: Cohort 2; FT-2102 (Single Agent): Participants with AML in morphologic complete remission (CR)/ complete remission with incomplete blood count recovery (CRi) after prior therapy with residual isocitrate dehydrogenase 1 ([IDH1]-R132 mutation were received single agent of FT-2102 150 mg BID in continuous 28-day cycles.
- Phase 2: Cohort 3; FT-2102 (Single Agent): Participants with R/R AML or MDS who were previously treated with FT-2102 and who underwent HSCT on-study then relapsed post-HSCT received single agent of FT-2102 150 mg BID in continuous 28-day cycles.
- Phase 2: Cohort 4; FT-2102 + Azacitidine (Combination Therapy): Participants with relapsed/refractory (R/R) AML that is naïve to prior hypomethylating therapy and IDH1 inhibitor therapy received combination therapy of azacitidine 75 mg/m^2 + FT-2102 150 mg BID in continuous 28-day cycles.
- Phase 2: Cohort 5; FT-2102 + Azacitidine (Combination Therapy): Participants with R/R AML/MDS that have inadequately responded to or have progressed on prior hypo-methylating therapy received combination therapy of azacitidine 75 mg/m^2 + FT-2102 150 mg BID in continuous 28-day cycles.
- Phase 2: Cohort 6; FT-2102 + Azacitidine (Combination Therapy): Participants with R/R AML/MDS that have been previously treated with single agent FT-2102 as their last therapy prior to study enrolment received combination therapy of azacitidine + FT-2102 150 mg BID in continuous 28-day cycles. Participants from the FT-2102 single agent cohorts of this study allowed to be enrolled in Cohort 6 after their disease progression.
- Phase 2: Cohort 7; FT-2102 (Single Agent): Participants who have not received any prior AML treatment but may have received a prior treatment for another hematologic malignancy be given single agent of FT-2102 150 mg BID in continuous 28-day cycles.
- Phase 2: Cohort 8; FT-2102 + Azacitidine (Combination Therapy): Participants who have not received any prior AML treatment but may have received a prior treatment for another hematologic malignancy be given combination therapy of azacitidine 75 mg/m^2 + FT-2102 150 mg BID in continuous 28-day cycles.
Period: Phase 1 (Dose Escalation)
Arm/Group | Phase 1: FT-2102 100mg QD (Single Agent; Dose Escalation) | Phase 1: FT-2102 150mg QD (Single Agent; Dose Escalation) | Phase 1: FT-2102 150mg BID (Single Agent; Dose Escalation) | Phase 1: FT-2102 300mg QD (Single Agent; Dose Escalation) | Phase 1: FT-2102 150mg QD+Azacitidine (Combination Therapy; Dose Escalation) | Phase 1: FT-2102 150mg BID+Azacitidine (Combination Therapy; Dose Escalation) | Phase 1: FT-2102 150mg BID (Single Agent; Dose Expansion) | Phase 1: FT-2102 150mg BID+Azacitidine (Combination Therapy; Dose Expansion) | Phase 1: FT-2102 150mg BID+ Cytarabine (Combination Therapy; Dose Expansion) | Phase 2: Cohort 1; FT-2102 (Single Agent) | Phase 2: Cohort 2; FT-2102 (Single Agent) | Phase 2: Cohort 3; FT-2102 (Single Agent) | Phase 2: Cohort 4; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 5; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 6; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 7; FT-2102 (Single Agent) | Phase 2: Cohort 8; FT-2102 + Azacitidine (Combination Therapy)
Started | 3 | 8 | 7 | 4 | 7 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 8 | 7 | 4 | 7 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 2 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 1 | 3 | 2 | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — HSCT Transplant | 0 | 1 | 2 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 1 (Dose Expansion)
Arm/Group | Phase 1: FT-2102 100mg QD (Single Agent; Dose Escalation) | Phase 1: FT-2102 150mg QD (Single Agent; Dose Escalation) | Phase 1: FT-2102 150mg BID (Single Agent; Dose Escalation) | Phase 1: FT-2102 300mg QD (Single Agent; Dose Escalation) | Phase 1: FT-2102 150mg QD+Azacitidine (Combination Therapy; Dose Escalation) | Phase 1: FT-2102 150mg BID+Azacitidine (Combination Therapy; Dose Escalation) | Phase 1: FT-2102 150mg BID (Single Agent; Dose Expansion) | Phase 1: FT-2102 150mg BID+Azacitidine (Combination Therapy; Dose Expansion) | Phase 1: FT-2102 150mg BID+ Cytarabine (Combination Therapy; Dose Expansion) | Phase 2: Cohort 1; FT-2102 (Single Agent) | Phase 2: Cohort 2; FT-2102 (Single Agent) | Phase 2: Cohort 3; FT-2102 (Single Agent) | Phase 2: Cohort 4; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 5; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 6; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 7; FT-2102 (Single Agent) | Phase 2: Cohort 8; FT-2102 + Azacitidine (Combination Therapy)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 31 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 31 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 10 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — HSCT Transplant | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1: FT-2102 100mg QD (Single Agent; Dose Escalation) | Phase 1: FT-2102 150mg QD (Single Agent; Dose Escalation) | Phase 1: FT-2102 150mg BID (Single Agent; Dose Escalation) | Phase 1: FT-2102 300mg QD (Single Agent; Dose Escalation) | Phase 1: FT-2102 150mg QD+Azacitidine (Combination Therapy; Dose Escalation) | Phase 1: FT-2102 150mg BID+Azacitidine (Combination Therapy; Dose Escalation) | Phase 1: FT-2102 150mg BID (Single Agent; Dose Expansion) | Phase 1: FT-2102 150mg BID+Azacitidine (Combination Therapy; Dose Expansion) | Phase 1: FT-2102 150mg BID+ Cytarabine (Combination Therapy; Dose Expansion) | Phase 2: Cohort 1; FT-2102 (Single Agent) | Phase 2: Cohort 2; FT-2102 (Single Agent) | Phase 2: Cohort 3; FT-2102 (Single Agent) | Phase 2: Cohort 4; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 5; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 6; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 7; FT-2102 (Single Agent) | Phase 2: Cohort 8; FT-2102 + Azacitidine (Combination Therapy)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 153 | 18 | 5 | 20 | 21 | 20 | 10 | 11
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 153 | 18 | 5 | 20 | 21 | 20 | 10 | 11
Not completed — Protocol Defined Disease Progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 65 | 8 | 2 | 4 | 9 | 11 | 3 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 27 | 0 | 1 | 1 | 1 | 2 | 2 | 3
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 7 | 0 | 5 | 7 | 0 | 1 | 4
Not completed — Transplant | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 2 | 0 | 6 | 1 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Not completed — Investigator Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 1 | 2 | 3 | 1 | 3 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all the participants who were enrolled in the study and have received at least one dose of FT-2102.
Groups:
- Phase 1: FT-2102 100mg QD (Single Agent; Dose Escalation): Participants with AML or MDS received single agent of FT-2102 100 mg orally QD in 28-day cycles until MTD or MED achieved.
- Phase 1: FT-2102 150mg BID+ Cytarabine (Combination Therapy; Dose Expansion): Participants with AML harboring IDH1 mutation received FT-2102 150 mg BID in combination with LDAC administered at the dose of 20 mg BID SC for 10 days every 28-day cycle until treatment discontinuation.
- Phase 2: Cohort 1; FT-2102 (Single Agent): Participants with R/R AML received single agent of FT-2102 150 mg BID in continuous 28-day cycles.
- Phase 2: Cohort 2; FT-2102 (Single Agent): Participants with AML in morphologic CR/CRi after prior therapy with residual IDH1-R132 mutation were received single agent of FT-2102 150 mg BID in continuous 28-day cycles.
- Phase 2: Cohort 4; FT-2102 + Azacitidine (Combination Therapy): Participants with R/R AML that is naïve to prior hypomethylating therapy and IDH1 inhibitor therapy received combination therapy of azacitidine 75 mg/m^2 + FT-2102 150 mg BID in continuous 28-day cycles.
- Total: Total of all reporting groups
Arm/Group | Phase 1: FT-2102 100mg QD (Single Agent; Dose Escalation) | Phase 1: FT-2102 150mg QD (Single Agent; Dose Escalation) | Phase 1: FT-2102 150mg BID (Single Agent; Dose Escalation) | Phase 1: FT-2102 300mg QD (Single Agent; Dose Escalation) | Phase 1: FT-2102 150mg QD+Azacitidine (Combination Therapy; Dose Escalation) | Phase 1: FT-2102 150mg BID+Azacitidine (Combination Therapy; Dose Escalation) | Phase 1: FT-2102 150mg BID (Single Agent; Dose Expansion) | Phase 1: FT-2102 150mg BID+Azacitidine (Combination Therapy; Dose Expansion) | Phase 1: FT-2102 150mg BID+ Cytarabine (Combination Therapy; Dose Expansion) | Phase 2: Cohort 1; FT-2102 (Single Agent) | Phase 2: Cohort 2; FT-2102 (Single Agent) | Phase 2: Cohort 3; FT-2102 (Single Agent) | Phase 2: Cohort 4; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 5; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 6; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 7; FT-2102 (Single Agent) | Phase 2: Cohort 8; FT-2102 + Azacitidine (Combination Therapy) | Total
Number analyzed (Participants) | 3 | 8 | 7 | 4 | 7 | 8 | 9 | 31 | 1 | 153 | 18 | 5 | 20 | 21 | 20 | 10 | 11 | 336
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 0 | 3 | 1 | 3 | 5 | 1 | 0 | 10 | 0 | 37 | 5 | 1 | 16 | 3 | 3 | 0 | 1 | 89
  65 - <75 years | 0 | 3 | 4 | 0 | 1 | 5 | 6 | 14 | 0 | 68 | 11 | 3 | 2 | 9 | 9 | 3 | 6 | 144
  >=75 years | 3 | 2 | 2 | 1 | 1 | 2 | 3 | 7 | 1 | 48 | 2 | 1 | 2 | 9 | 8 | 7 | 4 | 103
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 2 | 2 | 5 | 5 | 5 | 14 | 0 | 74 | 6 | 2 | 11 | 7 | 10 | 6 | 2 | 158
  Male | 1 | 3 | 5 | 2 | 2 | 3 | 4 | 17 | 1 | 79 | 12 | 3 | 9 | 14 | 10 | 4 | 9 | 178
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 5 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 5 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 15
  White | 3 | 5 | 7 | 2 | 6 | 6 | 8 | 19 | 1 | 71 | 10 | 4 | 11 | 14 | 13 | 5 | 6 | 191
  More than one race | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 16 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 7 | 0 | 56 | 7 | 0 | 8 | 4 | 7 | 5 | 3 | 99

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: A TEAE was defined as an adverse event (AE) that emerges during treatment, having been absent pre-treatment, or worsens relative to the pre-treatment state. An AE was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a product, whether or not considered related to the product. A serious adverse event (SAE) is defined as any untoward medical occurrence that at any dose results in death, or is life-threatening, or requires inpatient hospitalization or causes prolongation of existing hospitalization results in persistent or significant disability/incapacity, or may have caused a congenital anomaly/birth defect, or requires intervention to prevent permanent impairment or damage. Number of participants with TEAEs and SAEs is reported. Safety analysis set (SAS) included all the participants who have received at least one dose of study drug (FT-2102, azacitidine, or cytarabine).
Time Frame: Phase 1: From start of drug administration (Day 1) up to 28 days after last dose of study drug (up to 82 months)
Population: SAS analyzed. Since 150 mg BID has been established as MTD, the analysis was directed towards emphasizing findings that are most relevant for determining a safe and effective treatment strategy. Accordingly, data for the other dose levels (100 mg QD, 150 mg QD, and 300 mg QD) were combined as prespecified in statistical analysis plan (SAP).
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: FT-2102 (Single Agent): Participants with AML or MDS received single agent FT-2102 orally BID in 28-day cycles at dose levels of 150 mg until maximum MTD or maximum MED achieved.
- Phase 1: Total FT-2102 (Single Agent): Participants with AML or MDS received single agent FT-2102 orally QD and BID in 28-day cycles at the different dose levels (150 mg and ≤ 300 mg) until MTD or MED achieved.
- Phase 1: FT-2102 + Azacitidine (Combination Therapy): Participants with AML or MDS received combination therapy (FT-2102 + azacitidine 75 mg/m^2) orally BID in 28-day cycles at dose levels of 150 mg until MTD or MED achieved.
- Phase 1: Total FT-2102; FT-2102 + Azacitidine (Combination Therapy): Participants with AML or MDS received combination therapy (FT-2102 150 mg and ≤ 300 mg and azacitidine administered at the dose of 75 mg/m^2 for 7 days IV/SC per every 28-day cycle) until treatment discontinuation.
Arm/Group | Phase 1: FT-2102 (Single Agent) | Phase 1: Total FT-2102 (Single Agent) | Phase 1: FT-2102 + Azacitidine (Combination Therapy) | Phase 1: Total FT-2102; FT-2102 + Azacitidine (Combination Therapy)
Number analyzed (Participants) | 16 | 31 | 39 | 46
Participants
  TEAEs | 16 | 31 | 39 | 46
  SAEs | 10 | 23 | 30 | 36

2. Primary Outcome: Phase 1: Number of Participants With Change From Baseline in Clinically Significant Abnormal Laboratory Values
Description: Number of participants with change from baseline in clinically significant abnormal laboratory values for hematology, chemistry and coagulation with Grade <1 to 4 is reported. National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03 toxicity grade used to determine severity of AE. Grade 1: mild;asymptomatic/mild symptoms; Grade 2: moderate; minimal; Grade 3: severe/medically significant; Grade 4: life-threatening consequences, Grade 5: death.
Time Frame: Phase 1: From Baseline up to 28 days after last dose of study drug (up to 82 months)
Population: SAS analyzed. Since 150 mg BID has been established as MTD, the analysis was directed towards emphasizing findings that are most relevant for determining a safe and effective treatment strategy. Accordingly, data for the other dose levels (100 mg QD, 150 mg QD, and 300 mg QD) were combined as prespecified in SAP.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: Total FT-2102 (Single Agent): Participants with AML or MDS received single agent FT-2102 orally QD and BID in 28-day cycles at the differ-ent dose levels (150 mg and ≤ 300 mg) until MTD or MED achieved.
Arm/Group | Phase 1: FT-2102 (Single Agent) | Phase 1: Total FT-2102 (Single Agent) | Phase 1: FT-2102 + Azacitidine (Combination Therapy) | Phase 1: Total FT-2102; FT-2102 + Azacitidine (Combination Therapy)
Number analyzed (Participants) | 16 | 31 | 39 | 46
Participants
  Hematology: Hemoglobin; Increase(Grade <1) | 15 | 30 | 38 | 45
  Hematology: Hemoglobin; Increase (Grade 1) | 0 | 0 | 0 | 0
  Hematology: Hemoglobin; Increase (Grade 2) | 0 | 1 | 1 | 1
  Hematology: Hemoglobin; Increase (Grade 3) | 0 | 0 | 0 | 0
  Hematology: Hemoglobin; Increase (Grade 4) | 0 | 0 | 0 | 0
  Hematology: Hemoglobin; Increase (Grade 3 or 4) | 0 | 0 | 0 | 0
  Hematology: Hemoglobin; Decrease (Grade <1) | 0 | 0 | 0 | 0
  Hematology: Hemoglobin; Decrease (Grade 1) | 3 | 3 | 0 | 0
  Hematology: Hemoglobin; Decrease (Grade 2) | 1 | 7 | 9 | 10
  Hematology: Hemoglobin; Decrease (Grade 3) | 11 | 20 | 30 | 36
  Hematology: Hemoglobin; Decrease (Grade 4) | 0 | 0 | 0 | 0
  Hematology: Hemoglobin; Decrease(Grade 3 or 4) | 11 | 20 | 30 | 36
  Hematology: Platelets; Decrease (Grade <1) | 1 | 2 | 0 | 0
  Hematology: Platelets; Decrease (Grade 1) | 2 | 2 | 0 | 0
  Hematology: Platelets; Decrease (Grade 2) | 0 | 1 | 3 | 3
  Hematology: Platelets; Decrease (Grade 3) | 1 | 5 | 5 | 6
  Hematology: Platelets; Decrease (Grade 4) | 11 | 20 | 31 | 37
  Hematology: Platelets; Decrease (Grade 3 or 4) | 12 | 25 | 36 | 43
  Hematology: Leukocytes; Increase (Grade <1) | 14 | 28 | 36 | 43
  Hematology: Leukocytes; Increase (Grade 1) | 0 | 0 | 0 | 0
  Hematology: Leukocytes; Increase (Grade 2) | 0 | 0 | 0 | 0
  Hematology: Leukocytes; Increase (Grade 3) | 1 | 2 | 3 | 3
  Hematology: Leukocytes; Increase (Grade 4) | 0 | 0 | 0 | 0
  Hematology: Leukocytes; Increase (Grade 3 or 4) | 1 | 2 | 3 | 3
  Hematology: Leukocytes; Decrease (Grade <1) | 1 | 2 | 1 | 2
  Hematology: Leukocytes: Decrease (Grade 1) | 2 | 3 | 1 | 1
  Hematology: Leukocytes; Decrease (Grade 2) | 1 | 6 | 4 | 4
  Hematology: Leukocytes; Decrease (Grade 3) | 4 | 8 | 14 | 16
  Hematology: Leukocytes; Decrease (Grade 4) | 7 | 11 | 19 | 23
  Hematology: Leukocytes; Decrease (Grade 3 or 4) | 11 | 19 | 33 | 39
  Hematology: Neutrophils; Decrease (Grade <1) | 1 | 1 | 1 | 1
  Hematology: Neutrophils; Decrease (Grade 1) | 0 | 1 | 0 | 0
  Hematology: Neutrophils; Decrease (Grade 2) | 0 | 0 | 0 | 0
  Hematology: Neutrophils; Decrease (Grade 3) | 2 | 5 | 2 | 2
  Hematology: Neutrophils; Decrease (Grade 4) | 12 | 23 | 36 | 43
  Hematology: Neutrophils; Decrease (Grade 3 or 4) | 14 | 28 | 38 | 45
  Hematology: Lymphocytes; Increase (Grade <1) | 11 | 19 | 26 | 32
  Hematology: Lymphocytes; Increase (Grade 1) | 0 | 0 | 0 | 0
  Hematology: Lymphocytes; Increase (Grade 2) | 3 | 10 | 11 | 12
  Hematology: Lymphocytes: Increase (Grade 3) | 0 | 0 | 1 | 1
  Hematology: Lymphocytes; Increase (Grade 4) | 0 | 0 | 0 | 0
  Hematology: Lymphocytes; Increase (Grade 3 or 4) | 0 | 0 | 1 | 1
  Hematology: Lymphocytes; Decrease(Grade <1) | 1 | 3 | 2 | 2
  Hematology: Lymphocytes; Decrease(Grade 1) | 2 | 7 | 6 | 6
  Hematology: Lymphocytes; Decrease(Grade 2) | 5 | 6 | 10 | 14
  Hematology: Lymphocytes; Decrease(Grade 3) | 5 | 10 | 16 | 18
  Hematology: Lymphocytes; Decrease(Grade 4) | 1 | 3 | 4 | 5
  Hematology: Lymphocytes; Decrease(Grade 3 or 4) | 6 | 13 | 20 | 23
  Chemistry: Creatinine; Increase (Grade <1) | 0 | 3 | 2 | 3
  Chemistry: Creatinine; Increase (Grade 1) | 12 | 23 | 26 | 31
  Chemistry: Creatinine; Increase (Grade 2) | 3 | 4 | 10 | 11
  Chemistry: Creatinine; Increase (Grade 3) | 0 | 0 | 1 | 1
  Chemistry: Creatinine; Increase (Grade 4) | 0 | 0 | 0 | 0
  Chemistry: Creatinine; Increase (Grade 3 or 4) | 0 | 0 | 1 | 1
  Chemistry: Calcium; Increase (Grade <1) | 13 | 28 | 35 | 39
  Chemistry: Calcium; Increase (Grade 1) | 0 | 0 | 3 | 4
  Chemistry: Calcium; Increase (Grade 2) | 0 | 0 | 0 | 0
  Chemistry: Calcium; Increase (Grade 3) | 1 | 1 | 0 | 1
  Chemistry: Calcium; Increase (Grade 4) | 1 | 1 | 0 | 0
  Chemistry: Calcium; Increase (Grade 3 or 4) | 2 | 2 | 0 | 1
  Chemistry: Calcium; Decrease(Grade <1) | 6 | 12 | 13 | 16
  Chemistry: Calcium; Decrease(Grade 1) | 9 | 17 | 23 | 26
  Chemistry: Calcium; Decrease(Grade 2) | 0 | 1 | 1 | 1
  Chemistry: Calcium; Decrease(Grade 3) | 0 | 0 | 1 | 1
  Chemistry: Calcium; Decrease(Grade 4) | 0 | 0 | 0 | 0
  Chemistry: Calcium; Decrease(Grade 3 or 4) | 0 | 0 | 1 | 1
  Chemistry: Magnesium; Increase(Grade <1) | 15 | 28 | 33 | 40
  Chemistry: Magnesium; Increase(Grade 1) | 0 | 0 | 0 | 0
  Chemistry: Magnesium; Increase(Grade 2) | 0 | 0 | 0 | 0
  Chemistry: Magnesium; Increase(Grade 3) | 0 | 2 | 5 | 5
  Chemistry: Magnesium; Increase(Grade 4) | 0 | 0 | 0 | 0
  Chemistry: Magnesium; Increase(Grade 3 or 4) | 0 | 2 | 5 | 5
  Chemistry: Magnesium; Decrease(Grade <1) | 8 | 17 | 24 | 26
  Chemistry: Magnesium; Decrease(Grade 1) | 7 | 13 | 14 | 19
  Chemistry: Magnesium; Decrease(Grade 2) | 0 | 0 | 0 | 0
  Chemistry: Magnesium; Decrease(Grade 3) | 0 | 0 | 0 | 0
  Chemistry: Magnesium; Decrease(Grade 4) | 0 | 0 | 0 | 0
  Chemistry: Magnesium; Decrease(Grade 3 or 4) | 0 | 0 | 0 | 0
  Chemistry: Potassium; Increase(Grade <1) | 13 | 24 | 34 | 40
  Chemistry: Potassium; Increase(Grade 1) | 1 | 5 | 3 | 4
  Chemistry: Potassium; Increase(Grade 2) | 1 | 1 | 2 | 2
  Chemistry: Potassium; Increase(Grade 3) | 0 | 0 | 0 | 0
  Chemistry: Potassium; Increase(Grade 4) | 0 | 0 | 0 | 0
  Chemistry: Potassium; Increase(Grade 3 or 4) | 0 | 0 | 0 | 0
  Chemistry: Potassium; Decrease(Grade <1) | 10 | 16 | 21 | 23
  Chemistry: Potassium; Decrease(Grade 1) | 3 | 10 | 14 | 19
  Chemistry: Potassium; Decrease(Grade 2) | 0 | 0 | 0 | 0
  Chemistry: Potassium; Decrease(Grade 3) | 2 | 4 | 4 | 4
  Chemistry: Potassium; Decrease(Grade 4) | 0 | 0 | 0 | 0
  Chemistry: Potassium; Decrease (Grade 3 or 4) | 2 | 4 | 4 | 4
  Chemistry: Sodium; Increase (Grade <1) | 13 | 27 | 34 | 41
  Chemistry: Sodium; Increase (Grade 1) | 2 | 3 | 5 | 5
  Chemistry: Sodium; Increase (Grade 2) | 0 | 0 | 0 | 0
  Chemistry: Sodium; Increase (Grade 3) | 0 | 0 | 0 | 0
  Chemistry: Sodium; Increase (Grade 4) | 0 | 0 | 0 | 0
  Chemistry: Sodium; Increase (Grade 3 or 4) | 0 | 0 | 0 | 0
  Chemistry: Sodium; Decrease (Grade <1) | 7 | 15 | 17 | 19
  Chemistry: Sodium; Decrease (Grade 1) | 7 | 11 | 19 | 24
  Chemistry: Sodium; Decrease (Grade 2) | 0 | 0 | 0 | 0
  Chemistry: Sodium; Decrease (Grade 3) | 1 | 4 | 3 | 3
  Chemistry: Sodium; Decrease (Grade 4) | 0 | 0 | 0 | 0
  Chemistry: Sodium; Decrease (Grade 3 or 4) | 1 | 4 | 3 | 3
  Chemistry: Uric acid; Increase (Grade <1) | 10 | 21 | 25 | 31
  Chemistry: Uric acid; Increase (Grade 1) | 5 | 9 | 10 | 10
  Chemistry: Uric acid; Increase (Grade 2) | 0 | 0 | 0 | 0
  Chemistry: Uric acid; Increase (Grade 3) | 0 | 0 | 0 | 0
  Chemistry: Uric acid; Increase (Grade 4) | 0 | 0 | 3 | 4
  Chemistry: Uric acid; Increase (Grade 3 or 4) | 0 | 0 | 3 | 4
  Chemistry: Albumin; Decrease(Grade <1) | 6 | 12 | 14 | 16
  Chemistry: Albumin; Decrease(Grade 1) | 5 | 10 | 12 | 12
  Chemistry: Albumin; Decrease(Grade 2) | 2 | 6 | 12 | 16
  Chemistry: Albumin; Decrease(Grade 3) | 2 | 2 | 0 | 1
  Chemistry: Albumin; Decrease(Grade 4) | 0 | 0 | 0 | 0
  Chemistry: Albumin; Decrease(Grade 3 or 4) | 2 | 2 | 0 | 1
  Chemistry: Glucose; Increase (Grade <1) | 13 | 26 | 33 | 40
  Chemistry: Glucose; Increase (Grade 1) | 0 | 0 | 0 | 0
  Chemistry: Glucose; Increase (Grade 2) | 0 | 0 | 0 | 0
  Chemistry: Glucose; Increase (Grade 3) | 1 | 2 | 5 | 5
  Chemistry: Glucose; Increase (Grade 4) | 1 | 2 | 0 | 0
  Chemistry: Glucose; Increase (Grade 3 or 4) | 2 | 4 | 5 | 5
  Chemistry: Glucose; Decrease(Grade <1) | 14 | 29 | 32 | 39
  Chemistry: Glucose; Decrease(Grade 1) | 1 | 1 | 5 | 5
  Chemistry: Glucose; Decrease(Grade 2) | 0 | 0 | 1 | 1
  Chemistry: Glucose; Decrease(Grade 3) | 0 | 0 | 0 | 0
  Chemistry: Glucose; Decrease(Grade 4) | 0 | 0 | 0 | 0
  Chemistry: Glucose; Decrease(Grade 3 or 4) | 0 | 0 | 0 | 0
  Chemistry: Lipase; Increase (Grade <1) | 2 | 2 | 18 | 18
  Chemistry: Lipase; Increase (Grade 1) | 1 | 1 | 0 | 0
  Chemistry: Lipase; Increase (Grade 2) | 0 | 0 | 0 | 0
  Chemistry: Lipase; Increase (Grade 3) | 1 | 1 | 2 | 2
  Chemistry: Lipase; Increase (Grade 4) | 0 | 0 | 0 | 0
  Chemistry: Lipase; Increase (Grade 3 or 4) | 1 | 1 | 2 | 2
  Chemistry: Amylase; Decrease(Grade <1) | 4 | 5 | 19 | 19
  Chemistry: Amylase; Decrease(Grade 1) | 0 | 0 | 0 | 0
  Chemistry: Amylase; Decrease(Grade 2) | 0 | 0 | 0 | 0
  Chemistry: Amylase; Decrease(Grade 3) | 0 | 0 | 0 | 0
  Chemistry: Amylase; Decrease(Grade 4) | 0 | 0 | 0 | 0
  Chemistry: Amylase; Decrease(Grade 3 or 4) | 0 | 0 | 0 | 0
  Coagulation: Activated partial Thromboplastin Time; Increase(Grade <1) | 6 | 7 | 20 | 21
  Coagulation: Activated partial Thromboplastin Time; Increase(Grade 1) | 1 | 1 | 2 | 2
  Coagulation: Activated partial Thromboplastin Time; Increase(Grade 2) | 0 | 0 | 1 | 1
  Coagulation: Activated partial Thromboplastin Time; Increase(Grade 3) | 0 | 0 | 1 | 1
  Coagulation: Activated partial Thromboplastin Time; Increase(Grade 4) | 0 | 0 | 0 | 0
  Coagulation: Activated partial Thromboplastin Time; Increase (Grade 3 or 4) | 0 | 0 | 1 | 1

3. Primary Outcome: Phase 1: Number of Participants With Change From Baseline in Clinically Significant Abnormal Electrocardiogram (ECG)
Description: Number of participants with change from baseline in clinically significant abnormal ECG parameter (QTcF) is reported. QT interval was the time between the start of the Q wave and the end of the T wave in the cardiac electrical cycle. QTcF was the QT interval corrected for heart rate using Fridericia's formula: QTcF = QT divided by cube root of 60/heart rate.
Time Frame: Phase 1: From Baseline up to 28 days after last dose of study drug (up to 82 months)
Population: SAS. Here, N=Number of participants with available data. Since 150mg BID has been established as MTD, analysis was directed towards emphasizing findings that are most relevant for determining safe and effective treatment strategy. Accordingly, data for other dose levels (100mg QD, 150mg QD, and 300mg QD) were combined as prespecified in SAP.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: FT-2102 (Single Agent) | Phase 1: Total FT-2102 (Single Agent) | Phase 1: FT-2102 + Azacitidine (Combination Therapy) | Phase 1: Total FT-2102; FT-2102 + Azacitidine (Combination Therapy)
Number analyzed (Participants) | 15 | 30 | 38 | 45
Participants
  <=450 msec | 10 | 16 | 23 | 26
  >450 to <=480 msec | 4 | 11 | 10 | 13
  >480 to <=500 msec | 0 | 2 | 1 | 2
  >500 msec | 1 | 1 | 4 | 4
  >30 to <=60 msec | 2 | 8 | 13 | 14
  >60 msec | 1 | 2 | 5 | 6

4. Primary Outcome: Phase 2, Cohort 1: Percentage of Participants With Complete Remission (CR) Plus Complete Remission With Partial Hematological Recovery (CRh) for Acute Myeloid Leukemia Assessed by Investigator Based on International Working Group (IWG) Response Criteria
Description: Percentage of participants with CR plus CRh (CR, Molecular CR [CRm], Cytogenetic CR [CRc], CRh) is re-ported. CR is defined as bone marrow blasts less than (<) 5 percent (%) (in aspirate with spicules and 200 nucleated cells), no blasts with auer rods, no extramedullary disease, absolute neutrophil count (ANC) greater than or equal to (>=) 1000/μL, platelet count >=100,000/μL and transfusion independ-ence. CRc is defined as CR with no residual cytogenetic abnormalities. CRm is defined as CR with unde-tectable IDH1m minimal residual disease (MRD) and CRh is defined as bone marrow blasts and partial recovery of peripheral blood counts (platelet count >50 × 10^9/L and ANC > 0.5 × 10^9/L).
Time Frame: Phase 2: up to 3 weeks post last dose of study drug or until the introduction of new anticancer therapy, whichever is earlier (up to 82 months)
Population: Efficacy evaluable analysis set included all participants in Phase 2, Cohort 1 with confirmed IDH1-R132 who have received the first dose of FT-2102 180 days or more prior to the analysis cutoff date. This outcome measure is applicable only for Cohort 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2: Cohort 1; FT-2102 (Single Agent)
Number analyzed (Participants) | 147
Percentage of participants | 35 [27.0 to 43.0]

5. Primary Outcome: Phase 2, Cohort 3, 4, 5, 6, 7, 8: Percentage of Participants With CR Plus CRh for Acute Myeloid Leukemia Assessed by Investigator Based on IWG Response Criteria
Description: Percentage of participants with CR plus CRh (CR, Molecular CR [CRm]), Cytogenetic CR [CRc], CRh) is re-ported. CR is defined as bone marrow blasts <5 % (in aspirate with spicules and 200 nucleated cells), no blasts with auer rods, no extramedullary disease, ANC >=1000/μL, platelet count >=100,000/μL and transfusion independ-ence. CRc is defined as CR with no residual cytogenetic abnormalities. CRm is de-fined as CR with undetectable IDH1m MRD and CRh is defined as bone marrow blasts and partial recovery of peripheral blood counts (platelet count >50 × 10^9/L and ANC > 0.5 × 10^9/L).
Time Frame: as for outcome 4
Population: FAS included all the participants who were enrolled in the study and have received at least one dose of FT-2102. This outcome measure is applicable for Cohort 3, 4, 5, 6, 7 and 8. Here, Overall Number of Participants Analyzed = participants with available data for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2: Cohort 3; FT-2102 (Single Agent) | Phase 2: Cohort 4; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 5; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 6; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 7; FT-2102 (Single Agent) | Phase 2: Cohort 8; FT-2102 + Azacitidine (Combination Therapy)
Number analyzed (Participants) | 5 | 19 | 13 | 20 | 10 | 11
Percentage of participants | 0 [0.0 to 52.2] | 47 [24.4 to 71.1] | 38 [13.9 to 68.4] | 30 [11.9 to 54.3] | 40 [12.2 to 73.8] | 45 [16.7 to 76.6]

6. Primary Outcome: Phase 2, Cohort 4 and 5: Percentage of Participants With CR for MDS Assessed by IWG Response Criteria
Description: Percentage of participants with complete remission (CR) is reported. CR is defined as bone marrow blast ≤ 5% myeloblasts with normal maturation of all cell lines, peripheral blood: Hgb ≥11 grams per deciliter (g/dL), platelets ≥ 100 × 10^9/L, neutrophils ≥ 1.0 × 10^9/L and blasts 0%.
Time Frame: as for outcome 4
Population: FAS included all the participants who were enrolled in the study and have received at least one dose of FT-2102. This outcome measure is applicable for Cohort 4 and 5. Here, Overall Number of Participants Analyzed = participants with available data for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2: Cohort 4; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 5; FT-2102 + Azacitidine (Combination Therapy)
Number analyzed (Participants) | 1 | 8
Percentage of participants | 0 [0.0 to 97.5] | 13 [0.3 to 52.7]

7. Primary Outcome: Phase 2, Cohort 2: Four-month Relapse Free Survival (RFS) Rate
Description: RFS is defined as the time between the date of first dose until relapse or death from any cause, whichever occurs first. RFS is calculated for all participants in Phase 2 Cohort 2. 4-Month RFS rate is defined as the percentage of participants in Phase 2 Cohort 2 who have not relapsed or died on or before their 4-month response evaluation.
Time Frame: Phase 2: From the date of first dose until relapse or death from any cause, whichever occurs first (up to 4 months)
Population: FAS included all the participants who were enrolled in the study and have received at least one dose of FT-2102. This outcome measure is applicable for Cohort 2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2: Cohort 2; FT-2102 (Single Agent)
Number analyzed (Participants) | 18
Percentage of participants | 83 [58.6 to 96.4]

8. Secondary Outcome: Phase 1: Area Under the Curve (AUClast) for FT-2102
Description: Area under the plasma concentration-time curve from zero time until the last measurable concentration is presented.
Time Frame: Phase 1: Cycle 1 Day 1 and Cycle 2 Day 1 (Cycle length= 28 days)
Population: The pharmacokinetic (PK) analysis set included those participants for whom it was possible to calculate at least 1 primary PK parameter and who had no major protocol deviations thought to influence the absorption, distribution, metabolism, and excretion of the FT-2102. Here, number anaylzed (n) = participants with available data for specific timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanograms per millilitre (h*ng/mL)
Groups:
- Phase 1: FT-2102 100 mg QD (Single Agent): Participants with AML or MDS received single agent FT-2102 orally QD in 28-day cycles at dose level of 100 mg until MTD or MED achieved.
- Phase 1: FT-2102 150 mg QD (Single Agent): Participants with AML or MDS received single agent FT-2102 orally QD in 28-day cycles at dose levels of 150 mg until MTD or MED achieved.
- Phase 1: FT-2102 300 mg QD (Single Agent): Participants with AML or MDS received single agent FT-2102 orally QD in 28-day cycles at dose levels of 300 mg until MTD or MED achieved.
- Phase 1: FT-2102 150 mg BID (Single Agent): Participants with AML or MDS received single agent FT-2102 orally BID in 28-day cycles at dose levels of 150 mg until MTD or MED achieved.
- Phase 1: FT-2102 150 mg QD+Azacitidine (Combination Therapy): Participants with AML or MDS received combination therapy (FT-2102 + azacitidine 75 mg/m^2) orally QD in 28-day cycles at dose levels of 150 mg until MTD or MED achieved
- Phase 1: FT-2102 150 mg BID+Azacitidine (Combination Therapy): Participants with AML or MDS received combination therapy (FT-2102 + azacitidine 75 mg/m^2) orally BID in 28-day cycles at dose levels of 150 mg until MTD or MED achieved.
Arm/Group | Phase 1: FT-2102 100 mg QD (Single Agent) | Phase 1: FT-2102 150 mg QD (Single Agent) | Phase 1: FT-2102 300 mg QD (Single Agent) | Phase 1: FT-2102 150 mg BID (Single Agent) | Phase 1: FT-2102 150 mg QD+Azacitidine (Combination Therapy) | Phase 1: FT-2102 150 mg BID+Azacitidine (Combination Therapy)
Number analyzed (Participants) | 3 | 8 | 4 | 6 | 7 | 8
Hour*nanograms per millilitre (h*ng/mL)
  Cycle 1 Day 1 | 5505 (146.9) | 8955 (63.7) | 12100 (75.4) | 2538 (34.2) | 8529 (51.1) | 2288 (71.7)
  Cycle 2 Day 1: number analyzed (Participants) | 3 | 5 | 4 | 6 | 6 | 5
  Cycle 2 Day 1 | 13080 (63.5) | 14130 (124.0) | 19140 (24.0) | 26360 (22.3) | 7468 (92.6) | 20640 (71.0)

9. Secondary Outcome: Phase 1: Maximum Plasma Concentration (Cmax) for FT-2102
Description: Maximum plasma concentration (Cmax) for FT-2102 is presented.
Time Frame: Phase 1: Cycle 1 Day 1 and Cycle 2 Day 1 (Cycle length= 28 days)
Population: The PK analysis set included those participants for whom it was possible to calculate at least 1 primary PK parameter and who had no major protocol deviations thought to influence the absorption, distribution, metabolism, and excretion of the FT-2102. Here, number anaylzed (n) = participants with available data for specific timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per millilitre (ng/mL)
Groups:
- Phase: FT-2102 150 mg BID (Single Agent): Participants with AML or MDS received single agent FT-2102 orally BID in 28-day cycles at dose levels of 150 mg until MTD or MED achieved.
Arm/Group | Phase 1: FT-2102 100 mg QD (Single Agent) | Phase 1: FT-2102 150 mg QD (Single Agent) | Phase 1: FT-2102 300 mg QD (Single Agent) | Phase: FT-2102 150 mg BID (Single Agent) | Phase 1: FT-2102 150 mg QD+Azacitidine (Combination Therapy) | Phase 1: FT-2102 150 mg BID+Azacitidine (Combination Therapy)
Number analyzed (Participants) | 3 | 8 | 4 | 6 | 7 | 8
Nanograms per millilitre (ng/mL)
  Cycle 1 Day 1 | 571.5 (53.1) | 535.0 (58.7) | 708.0 (58.2) | 495.5 (37.4) | 543.3 (39.8) | 439.9 (56.2)
  Cycle 2 Day 1: number analyzed (Participants) | 3 | 5 | 4 | 6 | 6 | 5
  Cycle 2 Day 1 | 1913 (47.9) | 1998 (112.9) | 2907 (36.1) | 3703 (20.8) | 1101 (75.4) | 3183 (51.5)

10. Secondary Outcome: Phase 1: Time to Maximum Plasma Concentration (Tmax) for FT-2102
Description: Time to reach the maximum plasma concentration (Tmax) is presented.
Time Frame: Phase 1: Cycle 1 Day 1 and Cycle 2 Day 1 (Cycle length= 28 days)
Population: as for outcome 9
Measure: Median (Full Range); unit: hour
Arm/Group | Phase 1: FT-2102 100 mg QD (Single Agent) | Phase 1: FT-2102 150 mg QD (Single Agent) | Phase 1: FT-2102 300 mg QD (Single Agent) | Phase 1: FT-2102 150 mg BID (Single Agent) | Phase 1: FT-2102 150 mg QD+Azacitidine (Combination Therapy) | Phase 1: FT-2102 150 mg BID+Azacitidine (Combination Therapy)
Number analyzed (Participants) | 3 | 8 | 4 | 6 | 7 | 8
hour
  Cycle 1 Day 1 | 4.05 [2.22 to 4.12] | 4.00 [2.02 to 24.00] | 23.83 [4.00 to 24.00] | 5.79 [1.00 to 7.83] | 4.02 [2.00 to 22.55] | 3.13 [2.03 to 4.12]
  Cycle 2 Day 1: number analyzed (Participants) | 3 | 5 | 4 | 6 | 6 | 5
  Cycle 2 Day 1 | 2.23 [2.13 to 4.00] | 2.00 [1.00 to 2.12] | 1.00 [0.00 to 1.08] | 3.00 [0.00 to 7.50] | 2.29 [2.00 to 4.00] | 1.18 [0.00 to 2.07]

11. Secondary Outcome: Phase 1: Time to Response (TTR) for AML
Description: TTR is the time in months between the first dose of study drug and documentation of the first overall response for participants who achieve a PR or better. This analysis was performed only on participants who have achieved PR or better as a best overall response.
Time Frame: Phase 1: Time from first dose of study drug until documentation of the first overall response (up to 82 months)
Population: FAS. N=participants with PR or better as best overall response. Since 150mg BID has been established as MTD, analysis was directed towards emphasizing findings that are most relevant for determining safe and effective treatment strategy. Accordingly, data for other dose levels (100mg QD, 150mg QD, and 300mg QD) were combined as prespecified in SAP.
Measure: Median (Full Range); unit: Months
Arm/Group | Phase 1: FT-2102 (Single Agent) | Phase 1: Total FT-2102 (Single Agent) | Phase 1: FT-2102 + Azacitidine (Combination Therapy) | Phase 1: Total FT-2102; FT-2102 + Azacitidine (Combination Therapy)
Number analyzed (Participants) | 5 | 10 | 18 | 22
Months | 1.90 [1.0 to 2.9] | 1.90 [1.0 to 4.7] | 1.90 [1.0 to 5.6] | 1.90 [1.0 to 5.6]

12. Secondary Outcome: Phase 1: Duration of Overall Response for AML
Description: Duration of response is defined as the time from the date of the first response to the date of the relapse or death. The estimation of median duration of overall response was done by Kaplan-Meier method.
Time Frame: Phase 1: From date of the first response to the date of the relapse or death (up to 82 months)
Population: FAS. N=participants with available data for this outcome measure. Since 150mg BID has been established as MTD, analysis was directed towards emphasizing findings that are most relevant for determining safe and effective treatment strategy. Accordingly, data for other dose levels(100mg QD, 150mg QD, and 300mg QD)were combined as prespecified in SAP.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1: FT-2102 (Single Agent) | Phase 1: Total FT-2102 (Single Agent) | Phase 1: FT-2102 + Azacitidine (Combination Therapy) | Phase 1: Total FT-2102; FT-2102 + Azacitidine (Combination Therapy)
Number analyzed (Participants) | 5 | 10 | 18 | 22
Months | 3.60 [1.70 to NA] — Since the upper confidence limits for the survivor function lies above 0.5, it is not possible to estimate the upper confidence limit for the median. | 2.90 [0.90 to 6.40] | 22.00 [3.20 to NA] — Since the upper confidence limits for the survivor function lies above 0.5, it is not possible to estimate the upper confidence limit for the median. | 22.00 [3.20 to NA] — Since the upper confidence limits for the survivor function lies above 0.5, it is not possible to estimate the upper confidence limit for the median.

13. Secondary Outcome: Phase 1: Time to Response (TTR ) for MDS
Description: as for outcome 11
Time Frame: Phase 1: Time from first dose of study drug until documentation of the first overall response (up to 82 months)
Population: FAS. N=participants with PR or better as best overall response. Since 150mg BID has been established as MTD, analysis was directed towards emphasizing findings that are most relevant for determining safe and effective treatment strategy. Accordingly, data for other dose levels(100mg QD, 150mg QD, and 300mg QD) were combined as prespecified in SAP.
Measure: Median (Full Range); unit: Months
Arm/Group | Phase 1: FT-2102 (Single Agent) | Phase 1: Total FT-2102 (Single Agent) | Phase 1: FT-2102 + Azacitidine (Combination Therapy) | Phase 1: Total FT-2102; FT-2102 + Azacitidine (Combination Therapy)
Number analyzed (Participants) | 2 | 2 | 6 | 6
Months | 4.65 [1.0 to 8.3] | 4.65 [1.0 to 8.3] | 2.20 [1.0 to 8.5] | 2.20 [1.0 to 8.5]

14. Secondary Outcome: Phase 2: Time to Response (TTR) for Acute Myeloid Leukemia (AML)
Description: as for outcome 11
Time Frame: Phase 2: Time from first dose of study drug until documentation of the first overall response (up to 82 months)
Population: FAS included all the participants who were enrolled in the study and have received at least one dose of FT-2102. Here, Overall Number of Participants Analyzed = participants with PR or better as a best overall response. Data is reported only for Cohort 1, 3, 4, 5, 6, 7 and 8.
Measure: Median (Full Range); unit: Months
Arm/Group | Phase 2: Cohort 1; FT-2102 (Single Agent) | Phase 2: Cohort 3; FT-2102 (Single Agent) | Phase 2: Cohort 4; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 5; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 6; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 7; FT-2102 (Single Agent) | Phase 2: Cohort 8; FT-2102 + Azacitidine (Combination Therapy)
Number analyzed (Participants) | 75 | 0 | 13 | 6 | 8 | 5 | 7
Months | 1.90 [0.9 to 10.2] |  | 1.80 [0.9 to 3.8] | 2.50 [1.0 to 4.2] | 2.50 [1.0 to 7.6] | 1.90 [1.8 to 3.9] | 2.80 [1.1 to 5.6]

15. Secondary Outcome: Phase 2: Duration of Overall Response for Acute Myeloid Leukemia (AML)
Description: Duration of overall response is defined as the time from the date of the first response to the date of the relapse or death. The estimation of median duration of overall response was done by Kaplan-Meier method.
Time Frame: Phase 2: From the date of the first response to the date of the relapse or death (up to 82 months)
Population: FAS included all the participants who were enrolled in the study and have received at least one dose of FT-2102. Data is reported only for Cohort 1, 4, 5, 6, 7 and 8. No participants achieved an overall response in Phase 2 Cohort 3. Duration of Response is not calculated for Phase 2 Cohort 2. Here, Overall Number of Participants Analyzed = participants with overall response for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: Cohort 1; FT-2102 (Single Agent) | Phase 2: Cohort 4; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 5; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 6; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 7; FT-2102 (Single Agent) | Phase 2: Cohort 8; FT-2102 + Azacitidine (Combination Therapy)
Number analyzed (Participants) | 75 | 13 | 6 | 8 | 5 | 7
Months | 14.80 [7.40 to 19.40] | 20.00 [1.90 to 28.80] | 7.25 [4.90 to NA] — Since the upper confidence limits for the survivor function lies above 0.5, it is not possible to estimate the upper confidence limit for the median. | 4.65 [2.80 to NA] — Since the upper confidence limits for the survivor function lies above 0.5, it is not possible to estimate the upper confidence limit for the median. | 10.60 [3.5 to 39.6] | 20.90 [5.60 to NA] — Since the upper confidence limits for the survivor function lies above 0.5, it is not possible to estimate the upper confidence limit for the median.

16. Secondary Outcome: Phase 2, Cohort 4 and Cohort 5: Time to Response (TTR) for Myelodysplastic Syndrome (MDS)
Description: as for outcome 11
Time Frame: Phase 2: Time from first dose of study drug until documentation of the first overall response (up to 82 months)
Population: FAS included all the participants who were enrolled in the study and have received at least one dose of FT-2102. This outcome measure is applicable for Cohort 4 and 5. Here, Overall Number of Participants Analyzed = participants with PR or better as a best overall response.
Measure: Median (Full Range); unit: Months
Arm/Group | Phase 2: Cohort 4; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 5; FT-2102 + Azacitidine (Combination Therapy)
Number analyzed (Participants) | 1 | 4
Months | 3.30 [3.3 to 3.3] | 1.50 [1.0 to 13.0]

17. Secondary Outcome: Phase 2, Cohort 4 and Cohort 5: Duration of Overall Response for Myelodysplastic Syndrome (MDS)
Description: Duration of overall response was calculated similarly to DCR but was assessed the time in months between documentation of the first response of PR or better until the date of relapse, death, whichever is earlier. The estimation of median duration of overall response was done by Kaplan-Meier method. The median duration of overall response is defined as the time at which 50% of the participants in a study have experienced the event of interest (relapse or death). Given the presence of only a single participant in the sample, there is an absence of variability in outcomes, and therefore, it was not possible to ascertain a time point at which half of the participants have experienced the event. Hence, median value could not be calculated.
Time Frame: Phase 2: From the documentation of the first response of PR or better until the date of relapse, death, whichever is earlier (up to 82 months)
Population: FAS included all the participants who were enrolled in the study and have received at least one dose of FT-2102. This outcome measure is applicable only for cohort 4 and 5. Here, Overall Number of Participants Analyzed = participants with overall response for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: Cohort 4; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 5; FT-2102 + Azacitidine (Combination Therapy)
Number analyzed (Participants) | 1 | 4
Months | NA [NA to NA] — Median and 95% CI could not be calculated since there is only one participant for Cohort 4. | 11.90 [2.80 to NA] — Since the upper confidence limits for the survivor function lies above 0.5, it is not possible to estimate the upper confidence limit for the median for Cohort 5.

18. Secondary Outcome: Phase 2, Cohort 2: Time to Relapse-Free Survival (RFS)
Description: RFS was calculated for all participants in Phase 2 Cohort 2. RFS is defined as the time (in months) between the date of first dose until relapse or death from any cause, whichever occurs first. Relapse free survival time to event is reported for all participants in Cohort 2.
Time Frame: Phase 2: From the date of first dose until relapse or death from any cause, whichever occurs first (up to 82 months)
Population: Full analysis set (FAS) included all the participants who were enrolled in the study and have received at least one dose of FT-2102. This outcome measure is applicable for Cohort 2.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: Cohort 2; FT-2102 (Single Agent)
Number analyzed (Participants) | 18
Months | 18.40 [9.50 to NA] — Since the upper confidence limits for the survivor function lies above 0.5, it is not possible to estimate the upper confidence limit for the median.

19. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: OS is defined as the time in months from the first dose of study drug until death from any cause. For the participants who are not known to have died by the end of study follow-up, OS will be censored on the date the participants was last known to be alive. OS is calculated using Kaplan-Meier method.
Time Frame: Phase 2: From first dose of study drug until death from any cause (up to 82 months)
Population: FAS included all the participants who were enrolled in the study and have received at least one dose of FT-2102.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: Cohort 1; FT-2102 (Single Agent) | Phase 2: Cohort 2; FT-2102 (Single Agent) | Phase 2: Cohort 3; FT-2102 (Single Agent) | Phase 2: Cohort 4; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 5; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 6; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 7; FT-2102 (Single Agent) | Phase 2: Cohort 8; FT-2102 + Azacitidine (Combination Therapy)
Number analyzed (Participants) | 153 | 18 | 5 | 20 | 21 | 20 | 10 | 11
Months | 11.60 [8.90 to 15.50] | NA [27.30 to NA] — The median was not reached, since more than half of the participants in the study had not experienced the event of death at the time of analysis. | 1.20 [1.10 to NA] — Since the upper confidence limits for the survivor function lies above 0.5, it is not possible to estimate the upper confidence limit for the median. | 25.20 [13.60 to NA] — Since the upper confidence limits for the survivor function lies above 0.5, it is not possible to estimate the upper confidence limit for the median. | 11.60 [5.00 to 27.50] | 10.20 [4.40 to 17.90] | 14.00 [1.00 to 19.10] | 18.70 [1.60 to NA] — Since the upper confidence limits for the survivor function lies above 0.5, it is not possible to estimate the upper confidence limit for the median.

20. Secondary Outcome: Phase 2: Event-free Survival (EFS)
Description: EFS is defined as the time in months between first dose of study drug and disease progression, relapse, death from any cause, treatment failure, or start of other (non-protocol study drug) new antileukemia therapy, whichever occurs first.
Time Frame: Phase 2: From first dose of study drug to disease progression, relapse, death from any cause, treatment failure, or start of other (non-protocol study drug) new antileukemia therapy (up to 82 months)
Population: FAS included all the participants who were enrolled in the study and have received at least one dose of FT-2102
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: Cohort 1; FT-2102 (Single Agent) | Phase 2: Cohort 2; FT-2102 (Single Agent) | Phase 2: Cohort 3; FT-2102 (Single Agent) | Phase 2: Cohort 4; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 5; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 6; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 7; FT-2102 (Single Agent) | Phase 2: Cohort 8; FT-2102 + Azacitidine (Combination Therapy)
Number analyzed (Participants) | 153 | 18 | 5 | 20 | 21 | 20 | 10 | 11
Months | 5.50 [4.30 to 7.40] | 18.40 [9.50 to NA] — Since the upper confidence limits for the survivor function lies above 0.5, it is not possible to estimate the upper confidence limit for the median. | 1.05 [0.80 to NA] — Since the upper confidence limits for the survivor function lies above 0.5, it is not possible to estimate the upper confidence limit for the median. | 5.70 [1.90 to 16.40] | 7.80 [2.10 to 10.20] | 4.80 [2.50 to 9.70] | 5.50 [0.30 to NA] — Since the upper confidence limits for the survivor function lies above 0.5, it is not possible to estimate the upper confidence limit for the median. | 8.10 [1.60 to 33.00]

21. Secondary Outcome: Phase 2: Transfusion Independence
Description: Transfusion independence is defined as the number of participants who experience at least a 56-day period during any point on treatment without requiring a transfusion of RBC and/or platelet transfusion. Participants are classified as either "dependent" or "independent" at baseline based on their transfusion history. Those who received either platelets or pRBC or both within 8 weeks prior to the first dose of FT-2102 are considered "dependent". Number of participants with transfusion independent is reported here.
Time Frame: Phase 2: From baseline (8 weeks prior to first dose) up to treatment period (up to 82 months)
Population: FAS included all the participants who were enrolled in the study and have received at least one dose of FT-2102.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Cohort 1; FT-2102 (Single Agent) | Phase 2: Cohort 2; FT-2102 (Single Agent) | Phase 2: Cohort 3; FT-2102 (Single Agent) | Phase 2: Cohort 4; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 5; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 6; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 7; FT-2102 (Single Agent) | Phase 2: Cohort 8; FT-2102 + Azacitidine (Combination Therapy)
Number analyzed (Participants) | 153 | 18 | 5 | 20 | 21 | 20 | 10 | 11
Participants | 72 | 15 | 0 | 12 | 13 | 14 | 3 | 8

22. Secondary Outcome: Phase 2: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: A TEAE was defined as an AE that emerges during treatment, having been absent pre-treatment, or worsens relative to the pre-treatment state. An AE was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a product, whether or not considered related to the product. A SAE is defined as any untoward medical occur-rence that at any dose results in death, or is life-threatening, or requires inpatient hospitalization or causes prolongation of existing hospitalization results in persistent or significant disability/incapacity, or may have caused a congenital anomaly/birth defect, or requires intervention to prevent permanent impairment or damage. Number of participants with TEAEs and SAEs is reported.
Time Frame: Phase 2: From start of drug administration (Day 1) up to 28 days after last dose of study drug (up to 82 months)
Population: Safety analysis set included all the participants who have received at least one dose of study drug (FT-2102, azacitidine, or cytarabine).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Cohort 1; FT-2102 (Single Agent) | Phase 2: Cohort 2; FT-2102 (Single Agent) | Phase 2: Cohort 3; FT-2102 (Single Agent) | Phase 2: Cohort 4; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 5; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 6; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 7; FT-2102 (Single Agent) | Phase 2: Cohort 8; FT-2102 + Azacitidine (Combination Therapy)
Number analyzed (Participants) | 153 | 18 | 5 | 20 | 21 | 20 | 10 | 11
Participants
  TEAEs | 153 | 18 | 5 | 19 | 21 | 19 | 10 | 11
  SAEs | 115 | 6 | 4 | 12 | 18 | 13 | 8 | 9

23. Secondary Outcome: Phase 2: Number of Participants With Change From Baseline in Clinically Significant Abnormal Laboratory Values
Description: as for outcome 2
Time Frame: Phase 2: From Baseline up to 28 days after last dose of study drug (up to 82 months)
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2: Cohort 2; FT-2102 (Single Agent): Participants with AML in morphologic CR)/CRi after prior therapy with residual IDH1-R132 mutation were received single agent of FT-2102 150 mg BID in continuous 28-day cycles.
Arm/Group | Phase 2: Cohort 1; FT-2102 (Single Agent) | Phase 2: Cohort 2; FT-2102 (Single Agent) | Phase 2: Cohort 3; FT-2102 (Single Agent) | Phase 2: Cohort 4; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 5; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 6; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 7; FT-2102 (Single Agent) | Phase 2: Cohort 8; FT-2102 + Azacitidine (Combination Therapy)
Number analyzed (Participants) | 153 | 18 | 5 | 20 | 21 | 20 | 10 | 11
Participants
  Hematology: Hemoglobin; Increase (Grade <1) | 146 | 18 | 5 | 19 | 20 | 20 | 10 | 10
  Hematology: Hemoglobin; Increase (Grade 1) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Hematology: Hemoglobin; Increase (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hematology: Hemoglobin; Increase (Grade 3) | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hematology: Hemoglobin; Increase (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hematology: Hemoglobin; Increase (Grade 3 or 4) | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hematology: Hemoglobin; Decrease (Grade <1) | 3 | 3 | 0 | 0 | 0 | 1 | 0 | 0
  Hematology: Hemoglobin; Decrease (Grade 1) | 17 | 8 | 0 | 1 | 0 | 2 | 1 | 0
  Hematology: Hemoglobin; Decrease (Grade 2) | 46 | 3 | 1 | 7 | 3 | 5 | 2 | 2
  Hematology: Hemoglobin; Decrease (Grade 3) | 86 | 4 | 4 | 11 | 18 | 12 | 7 | 9
  Hematology: Hemoglobin; Decrease (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hematology: Hemoglobin; Decrease (Grade 3 or 4) | 86 | 4 | 4 | 11 | 18 | 12 | 7 | 9
  Hematology: Platelets; Decrease (Grade <1) | 3 | 3 | 0 | 0 | 0 | 0 | 1 | 0
  Hematology: Platelets; Decrease (Grade 1) | 19 | 8 | 0 | 1 | 0 | 3 | 0 | 0
  Hematology: Platelets; Decrease (Grade 2) | 14 | 3 | 0 | 2 | 1 | 1 | 0 | 2
  Hematology: Platelets; Decrease (Grade 3) | 25 | 3 | 1 | 3 | 2 | 5 | 2 | 3
  Hematology: Platelets; Decrease (Grade 4) | 91 | 1 | 4 | 13 | 18 | 11 | 7 | 6
  Hematology: Platelets; Decrease (Grade 3 or 4) | 116 | 4 | 5 | 16 | 20 | 16 | 9 | 9
  Hematology: Leukocytes; Increase (Grade <1) | 150 | 18 | 5 | 18 | 20 | 19 | 10 | 11
  Hematology: Leukocytes; Increase (Grade 1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hematology: Leukocytes; Increase (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hematology: Leukocytes; Increase (Grade 3) | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 0
  Hematology: Leukocytes; Increase (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hematology: Leukocytes; Increase (Grade 3 or 4) | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 0
  Hematology: Leukocytes; Decrease (Grade <1) | 17 | 1 | 2 | 0 | 2 | 2 | 3 | 0
  Hematology: Leukocytes; Decrease (Grade 1) | 8 | 2 | 0 | 0 | 1 | 3 | 0 | 0
  Hematology: Leukocytes; Decrease (Grade 2) | 20 | 7 | 0 | 3 | 0 | 0 | 2 | 0
  Hematology: Leukocytes; Decrease (Grade 3) | 50 | 6 | 1 | 4 | 6 | 5 | 3 | 4
  Hematology: Leukocytes; Decrease (Grade 4) | 57 | 2 | 2 | 12 | 12 | 10 | 2 | 7
  Hematology: Leukocytes; Decrease (Grade 3 or 4) | 107 | 8 | 3 | 16 | 18 | 15 | 5 | 11
  Hematology: Neutrophils; Decrease (Grade <1) | 1 | 2 | 0 | 1 | 0 | 3 | 1 | 0
  Hematology: Neutrophils; Decrease (Grade 1) | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Hematology: Neutrophils; Decrease (Grade 2) | 6 | 5 | 0 | 0 | 0 | 0 | 1 | 0
  Hematology: Neutrophils; Decrease (Grade 3) | 21 | 4 | 0 | 1 | 1 | 1 | 2 | 0
  Hematology: Neutrophils; Decrease (Grade 4) | 117 | 6 | 5 | 17 | 19 | 15 | 6 | 10
  Hematology: Neutrophils; Decrease (Grade 3 or 4) | 138 | 10 | 5 | 18 | 20 | 16 | 8 | 10
  Hematology: Lymphocytes; Increase (Grade <1) | 103 | 17 | 2 | 14 | 19 | 14 | 8 | 8
  Hematology: Lymphocytes; Increase (Grade 1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hematology: Lymphocytes; Increase (Grade 2) | 36 | 1 | 3 | 5 | 1 | 4 | 2 | 1
  Hematology: Lymphocytes; Increase (Grade 3) | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Hematology: Lymphocytes; Increase (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hematology: Lymphocytes; Increase (Grade 3 or 4) | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Hematology: Lymphocytes; Decrease (Grade <1) | 18 | 2 | 1 | 1 | 1 | 1 | 1 | 1
  Hematology: Lymphocytes; Decrease (Grade 1) | 18 | 1 | 0 | 0 | 1 | 4 | 1 | 0
  Hematology: Lymphocytes; Decrease (Grade 2) | 36 | 7 | 0 | 7 | 4 | 4 | 3 | 3
  Hematology: Lymphocytes; Decrease (Grade 3) | 44 | 7 | 4 | 7 | 10 | 6 | 4 | 5
  Hematology: Lymphocytes; Decrease (Grade 4) | 27 | 1 | 0 | 4 | 5 | 3 | 1 | 0
  Hematology: Lymphocytes; Decrease (Grade 3 or 4) | 71 | 8 | 4 | 11 | 15 | 9 | 5 | 5
  Chemistry: Creatinine; Increase (Grade <1) | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  Chemistry: Creatinine; Increase (Grade 1) | 92 | 13 | 3 | 13 | 10 | 14 | 3 | 8
  Chemistry: Creatinine; Increase (Grade 2) | 55 | 4 | 1 | 5 | 10 | 6 | 6 | 3
  Chemistry: Creatinine; Increase (Grade 3) | 3 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Chemistry: Creatinine; Increase (Grade 4) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Chemistry: Creatinine; Increase (Grade 3 or 4) | 3 | 1 | 0 | 1 | 1 | 0 | 0 | 0
  Chemistry: Calcium; Increase (Grade <1) | 126 | 16 | 4 | 14 | 18 | 16 | 7 | 9
  Chemistry: Calcium; Increase (Grade 1) | 14 | 1 | 1 | 3 | 1 | 3 | 1 | 2
  Chemistry: Calcium; Increase (Grade 2) | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Chemistry: Calcium; Increase (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chemistry: Calcium; Increase (Grade 4) | 4 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Chemistry: Calcium; Increase (Grade 3 or 4) | 4 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Chemistry: Calcium; Decrease (Grade <1) | 83 | 13 | 4 | 14 | 13 | 16 | 4 | 6
  Chemistry: Calcium; Decrease (Grade 1) | 50 | 4 | 0 | 3 | 7 | 3 | 4 | 4
  Chemistry: Calcium; Decrease (Grade 2) | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Chemistry: Calcium; Decrease (Grade 3) | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0
  Chemistry: Calcium; Decrease (Grade 4) | 7 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Chemistry: Calcium; Decrease (Grade 3 or 4) | 9 | 0 | 1 | 1 | 0 | 1 | 0 | 1
  Chemistry: Magnesium; Increase (Grade <1) | 129 | 18 | 3 | 15 | 18 | 19 | 9 | 10
  Chemistry: Magnesium; Increase (Grade 1) | 13 | 0 | 2 | 1 | 3 | 1 | 0 | 1
  Chemistry: Magnesium; Increase (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chemistry: Magnesium; Increase (Grade 3) | 9 | 0 | 0 | 2 | 0 | 0 | 1 | 0
  Chemistry: Magnesium; Increase (Grade 4) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Chemistry: Magnesium; Increase (Grade 3 or 4) | 9 | 0 | 0 | 3 | 0 | 0 | 1 | 0
  Chemistry: Magnesium; Decrease (Grade <1) | 103 | 14 | 2 | 11 | 17 | 10 | 7 | 6
  Chemistry: Magnesium; Decrease (Grade 1) | 39 | 4 | 3 | 8 | 4 | 8 | 3 | 5
  Chemistry: Magnesium; Decrease (Grade 2) | 8 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Chemistry: Magnesium; Decrease (Grade 3) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chemistry: Magnesium; Decrease (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chemistry: Magnesium; Decrease (Grade 3 or 4) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chemistry: Potassium; Increase (Grade <1) | 120 | 12 | 5 | 17 | 16 | 16 | 7 | 9
  Chemistry: Potassium; Increase (Grade 1) | 28 | 4 | 0 | 2 | 4 | 2 | 3 | 2
  Chemistry: Potassium; Increase (Grade 2) | 4 | 2 | 0 | 0 | 1 | 2 | 0 | 0
  Chemistry: Potassium; Increase (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chemistry: Potassium; Increase (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chemistry: Potassium; Increase (Grade 3 or 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chemistry: Potassium; Decrease (Grade <1) | 73 | 14 | 1 | 7 | 16 | 12 | 6 | 5
  Chemistry: Potassium; Decrease (Grade 1) | 64 | 4 | 3 | 8 | 4 | 6 | 3 | 5
  Chemistry: Potassium; Decrease (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chemistry: Potassium; Decrease (Grade 3) | 9 | 0 | 0 | 4 | 1 | 2 | 1 | 1
  Chemistry: Potassium; Decrease (Grade 4) | 6 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Chemistry: Potassium; Decrease (Grade 3 or 4) | 15 | 0 | 1 | 4 | 1 | 2 | 1 | 1
  Chemistry: Sodium; Increase (Grade <1) | 139 | 17 | 4 | 18 | 19 | 20 | 9 | 8
  Chemistry: Sodium; Increase (Grade 1) | 13 | 0 | 0 | 1 | 2 | 0 | 1 | 3
  Chemistry: Sodium; Increase (Grade 2) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Chemistry: Sodium; Increase (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chemistry: Sodium; Increase (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chemistry: Sodium; Increase (Grade 3 or 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chemistry: Sodium; Decrease (Grade <1) | 77 | 15 | 3 | 13 | 13 | 12 | 5 | 5
  Chemistry: Sodium; Decrease (Grade 1) | 62 | 2 | 2 | 5 | 8 | 7 | 4 | 6
  Chemistry: Sodium; Decrease (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chemistry: Sodium; Decrease (Grade 3) | 12 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Chemistry: Sodium; Decrease (Grade 4) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Chemistry: Sodium; Decrease (Grade 3 or 4) | 13 | 1 | 0 | 1 | 0 | 1 | 1 | 0
  Chemistry: Uric acid; Increase (Grade <1) | 96 | 10 | 5 | 11 | 14 | 3 | 5 | 11
  Chemistry: Uric acid; Increase (Grade 1) | 49 | 8 | 0 | 6 | 5 | 6 | 4 | 0
  Chemistry: Uric acid; Increase (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chemistry: Uric acid; Increase (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chemistry: Uric acid; Increase (Grade 4) | 6 | 0 | 0 | 1 | 1 | 1 | 1 | 0
  Chemistry: Uric acid; Increase (Grade 3 or 4) | 6 | 0 | 0 | 1 | 1 | 1 | 1 | 0
  Chemistry: Albumin; Decrease (Grade <1) | 57 | 16 | 0 | 7 | 8 | 9 | 3 | 5
  Chemistry: Albumin; Decrease (Grade 1) | 41 | 1 | 2 | 6 | 7 | 6 | 2 | 2
  Chemistry: Albumin; Decrease (Grade 2) | 45 | 1 | 2 | 6 | 4 | 4 | 2 | 4
  Chemistry: Albumin; Decrease (Grade 3) | 8 | 0 | 1 | 0 | 2 | 1 | 3 | 0
  Chemistry: Albumin; Decrease (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chemistry: Albumin; Decrease (Grade 3 or 4) | 8 | 0 | 1 | 0 | 2 | 1 | 3 | 0
  Chemistry: Glucose; Increase (Grade <1) | 134 | 18 | 5 | 17 | 19 | 18 | 9 | 10
  Chemistry: Glucose; Increase (Grade 1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chemistry: Glucose; Increase (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chemistry: Glucose; Increase (Grade 3) | 16 | 0 | 0 | 2 | 1 | 2 | 1 | 1
  Chemistry: Glucose; Increase (Grade 4) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chemistry: Glucose; Increase (Grade 3 or 4) | 17 | 0 | 0 | 2 | 1 | 2 | 1 | 1
  Chemistry: Glucose; Decrease (Grade <1) | 136 | 15 | 5 | 17 | 18 | 19 | 10 | 10
  Chemistry: Glucose; Decrease (Grade 1) | 13 | 3 | 0 | 1 | 0 | 1 | 0 | 1
  Chemistry: Glucose; Decrease (Grade 2) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Chemistry: Glucose; Decrease (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chemistry: Glucose; Decrease (Grade 4) | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Chemistry: Glucose; Decrease (Grade 3 or 4) | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Chemistry: Lipase; Increase (Grade <1) | 108 | 8 | 5 | 12 | 16 | 17 | 8 | 7
  Chemistry: Lipase; Increase (Grade 1) | 13 | 4 | 0 | 3 | 5 | 1 | 0 | 3
  Chemistry: Lipase; Increase (Grade 2) | 12 | 3 | 0 | 2 | 0 | 1 | 1 | 0
  Chemistry: Lipase; Increase (Grade 3) | 11 | 1 | 0 | 0 | 0 | 1 | 1 | 0
  Chemistry: Lipase; Increase (Grade 4) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Chemistry: Lipase; Increase (Grade 3 or 4) | 12 | 1 | 0 | 0 | 0 | 1 | 0 | 1
  Chemistry: Amylase; Decrease (Grade <1) | 116 | 13 | 5 | 13 | 18 | 18 | 9 | 9
  Chemistry: Amylase; Decrease (Grade 1) | 24 | 3 | 0 | 3 | 2 | 0 | 1 | 1
  Chemistry: Amylase; Decrease (Grade 2) | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Chemistry: Amylase; Decrease (Grade 3) | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Chemistry: Amylase; Decrease (Grade 4) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Chemistry: Amylase; Decrease (Grade 3 or 4) | 5 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Coagulation: Activated partial Thromboplastin Time; Increase (Grade <1) | 82 | 14 | 0 | 13 | 13 | 8 | 4 | 5
  Coagulation: Activated partial Thromboplastin Time; Increase (Grade 1) | 15 | 0 | 1 | 0 | 3 | 2 | 0 | 3
  Coagulation: Activated partial Thromboplastin Time; Increase (Grade 2) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Coagulation: Activated partial Thromboplastin Time; Increase (Grade 3) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Coagulation: Activated partial Thromboplastin Time; Increase (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Coagulation: Activated partial Thromboplastin Time; Increase (Grade 3 or 4) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Phase 2: Number of Participants With Change From Baseline in Clinically Significant Abnormal Electrocardiogram (ECG)
Description: as for outcome 3
Time Frame: Phase 2: From Baseline up to 28 days after last dose of study drug (up to 82 months)
Population: Safety analysis set included all the participants who have received at least one dose of study drug (FT-2102, azacitidine, or cytarabine). Here, Overall Number of Participants Analyzed = participants with available data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Cohort 1; FT-2102 (Single Agent) | Phase 2: Cohort 2; FT-2102 (Single Agent) | Phase 2: Cohort 3; FT-2102 (Single Agent) | Phase 2: Cohort 4; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 5; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 6; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 7; FT-2102 (Single Agent) | Phase 2: Cohort 8; FT-2102 + Azacitidine (Combination Therapy)
Number analyzed (Participants) | 151 | 17 | 5 | 18 | 21 | 20 | 10 | 11
Participants
  <=450 msec | 90 | 11 | 1 | 9 | 9 | 11 | 9 | 4
  >450 to <=480 msec | 44 | 3 | 3 | 6 | 7 | 5 | 0 | 4
  >480 to <=500 msec | 12 | 1 | 1 | 1 | 2 | 1 | 1 | 1
  >500 msec | 5 | 2 | 0 | 2 | 3 | 3 | 0 | 2
  >30 to <=60 msec | 43 | 3 | 2 | 3 | 4 | 7 | 3 | 1
  >60 msec | 10 | 0 | 0 | 3 | 1 | 2 | 0 | 5

25. Secondary Outcome: Phase 2: Area Under the Curve (AUClast) for FT-2102
Description: Area under the plasma concentration-time curve from zero time until the last measurable concentration is presented.
Time Frame: Phase 2: Cycle 1 Day 1 and Cycle 2 Day 1 (Cycle length= 28 days)
Population: The PK analysis set included those participants for whom it was possible to calculate at least 1 primary PK parameter and who had no major protocol deviations thought to influence the absorption, distribution, metabolism, and excretion of the FT-2102. Here, Overall Number of Participants Analyzed (N) and number analyzed (n) = participants with available data for specific timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Phase 2: Cohort 1; FT-2102 150 mg BID (Single Agent): Participants with R/R AML received single agent of FT-2102 150 mg BID in continuous 28-day cycles.
- Phase 2: Cohort 2; FT-2102 150 mg BID (Single Agent): Participants with AML in morphologic CR/CRi after prior therapy with residual IDH1-R132 mutation were received single agent of FT-2102 150 mg BID in continuous 28-day cycles.
- Phase 2: Cohort 3; FT-2102 150 mg BID (Single Agent): Participants with R/R AML or MDS who were previously treated with FT-2102 and who underwent HSCT on-study then relapsed post-HSCT received single agent of FT-2102 150 mg BID in continuous 28-day cycles.
- Phase 2: Cohort 4; FT-2102 150 mg BID + Azacitidine (Combination Therapy): Participants with R/R AML that is naïve to prior hypomethylating therapy and IDH1 inhibitor therapy received combination therapy of azacitidine 75 mg/m^2 + FT-2102 150 mg BID in continuous 28-day cycles.
- Phase 2: Cohort 5; FT-2102 150 mg BID + Azacitidine (Combination Therapy): Participants with R/R AML/MDS that have inadequately responded to or have progressed on prior hypo-methylating therapy received combination therapy of azacitidine 75 mg/m^2 + FT-2102 150 mg BID in continuous 28-day cycles.
- Phase 2: Cohort 6; FT-2102 150 mg BID + Azacitidine (Combination Therapy): Participants with R/R AML/MDS that have been previously treated with single agent FT-2102 as their last therapy prior to study enrolment received combination therapy of azacitidine + FT-2102 150 mg BID in continuous 28-day cycles. Participants from the FT-2102 single agent cohorts of this study allowed to be enrolled in Cohort 6 after their disease progression.
- Phase 2: Cohort 7; FT-2102 150 mg BID (Single Agent): Participants who have not received any prior AML treatment but may have received a prior treatment for another hematologic malignancy be given single agent of FT-2102 150 mg BID in continuous 28-day cycles.
- Phase 2: Cohort 8; FT-2102 150 mg BID + Azacitidine (Combination Therapy): Participants who have not received any prior AML treatment but may have received a prior treatment for another hematologic malignancy be given combination therapy of azacitidine 75 mg/m^2 + FT-2102 150 mg BID in continuous 28-day cycles.
Arm/Group | Phase 2: Cohort 1; FT-2102 150 mg BID (Single Agent) | Phase 2: Cohort 2; FT-2102 150 mg BID (Single Agent) | Phase 2: Cohort 3; FT-2102 150 mg BID (Single Agent) | Phase 2: Cohort 4; FT-2102 150 mg BID + Azacitidine (Combination Therapy) | Phase 2: Cohort 5; FT-2102 150 mg BID + Azacitidine (Combination Therapy) | Phase 2: Cohort 6; FT-2102 150 mg BID + Azacitidine (Combination Therapy) | Phase 2: Cohort 7; FT-2102 150 mg BID (Single Agent) | Phase 2: Cohort 8; FT-2102 150 mg BID + Azacitidine (Combination Therapy)
Number analyzed (Participants) | 117 | 14 | 2 | 12 | 16 | 4 | 2 | 1
h*ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 117 | 14 | 2 | 12 | 16 | 3 | 2 | 1
  Cycle 1 Day 1 | 2836 (59.5) | 2657 (36.8) | 1880 (77.4) | 3051 (109.7) | 2031 (69.4) | 1701 (39.4) | 4165 (116.5) | 3898 (NA) — Geometric coefficient of variation could not be calculated due to small number of participants.
  Cycle 2 Day 1: number analyzed (Participants) | 88 | 12 | 0 | 11 | 14 | 4 | 1 | 1
  Cycle 2 Day 1 | 20610 (69.7) | 27710 (14.9) |  | 19820 (77.6) | 19610 (62.1) | 21810 (45.6) | 25880 (NA) — Geometric coefficient of variation could not be calculated due to small number of participants. | 19940 (NA) — Geometric coefficient of variation could not be calculated due to small number of participants.

26. Secondary Outcome: Phase 2: Maximum Plasma Concentration (Cmax) for FT-2102
Description: Maximum Plasma Concentartion (Cmax) for FT-2102 is presented.
Time Frame: Phase 2: Cycle 1 Day 1 and Cycle 2 Day 1 (Cycle length= 28 days)
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 2: Cohort 1; FT-2102 150 mg BID (Single Agent) | Phase 2: Cohort 2; FT-2102 150 mg BID (Single Agent) | Phase 2: Cohort 3; FT-2102 150 mg BID (Single Agent) | Phase 2: Cohort 4; FT-2102 150 mg BID + Azacitidine (Combination Therapy) | Phase 2: Cohort 5; FT-2102 150 mg BID + Azacitidine (Combination Therapy) | Phase 2: Cohort 6; FT-2102 150 mg BID + Azacitidine (Combination Therapy) | Phase 2: Cohort 7; FT-2102 150 mg BID (Single Agent) | Phase 2: Cohort 8; FT-2102 150 mg BID + Azacitidine (Combination Therapy)
Number analyzed (Participants) | 120 | 14 | 2 | 13 | 16 | 4 | 2 | 1
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 120 | 14 | 2 | 13 | 16 | 3 | 2 | 1
  Cycle 1 Day 1 | 534.5 (57.5) | 492.4 (29.3) | 388.8 (49.1) | 623.2 (75.8) | 404.1 (58.5) | 411.2 (9.0) | 747.5 (107.6) | 671 (NA) — Geometric coefficient of variation could not be calculated due to small number of participants.
  Cycle 2 Day 1: number analyzed (Participants) | 88 | 12 | 0 | 11 | 14 | 4 | 1 | 1
  Cycle 2 Day 1 | 3136 (62.0) | 3800 (14.7) |  | 3239 (68.7) | 2934 (53.6) | 3043 (39.3) | 3500 (NA) — Geometric coefficient of variation could not be calculated due to small number of participants. | 3080 (NA) — Geometric coefficient of variation could not be calculated due to small number of participants.

27. Secondary Outcome: Phase 2: Time to Maximum Plasma Concentration (Tmax) for FT-2102
Description: Time to reach the maximum plasma concentration (Tmax) for FT-2102 is presented.
Time Frame: Phase 2: Cycle 1 Day 1 and Cycle 2 Day 1 (Cycle length= 28 days)
Population: as for outcome 25
Measure: Median (Full Range); unit: hour
Arm/Group | Phase 2: Cohort 1; FT-2102 150 mg BID (Single Agent) | Phase 2: Cohort 2; FT-2102 150 mg BID (Single Agent) | Phase 2: Cohort 3; FT-2102 150 mg BID (Single Agent) | Phase 2: Cohort 4; FT-2102 150 mg BID + Azacitidine (Combination Therapy) | Phase 2: Cohort 5; FT-2102 150 mg BID + Azacitidine (Combination Therapy) | Phase 2: Cohort 6; FT-2102 150 mg BID + Azacitidine (Combination Therapy) | Phase 2: Cohort 7; FT-2102 150 mg BID (Single Agent) | Phase 2: Cohort 8; FT-2102 150 mg BID + Azacitidine (Combination Therapy)
Number analyzed (Participants) | 120 | 14 | 2 | 13 | 16 | 4 | 2 | 1
hour
  Cycle 1 Day 1: number analyzed (Participants) | 120 | 14 | 2 | 13 | 16 | 3 | 2 | 1
  Cycle 1 Day 1 | 4.00 [1.00 to 8.00] | 4.00 [2.00 to 8.00] | 5.00 [2.00 to 8.00] | 4.00 [2.00 to 8.00] | 4.00 [2.00 to 8.00] | 4.00 [2.00 to 8.00] | 3.00 [2.00 to 4.00] | 1.00 [1.00 to 1.00]
  Cycle 2 Day 1: number analyzed (Participants) | 88 | 12 | 0 | 11 | 14 | 4 | 1 | 1
  Cycle 2 Day 1 | 2.00 [0.00 to 8.00] | 1.00 [0.00 to 2.00] |  | 1.00 [0.00 to 8.00] | 1.00 [0.00 to 4.00] | 4.00 [0.00 to 8.00] | 0.00 [0 to 0] | 1.00 [1.00 to 1.00]

ADVERSE EVENTS:
Time Frame: From start of drug administration (Day 1) up to 28 days after last dose of study drug (up to 82 months)
Description: All presented AEs are TEAEs. TEAE is AE that emerges during treatment and absent pre-treatment/worsens relative to pre-treatment. 1 participant received FT-2102 with cytarabine, included in Phase 1 total column. Since 150mg BID has been established as MTD, analysis was directed towards emphasizing findings that are most relevant for determining safe and effective treatment strategy. Accordingly, data for other dose levels(100mg QD, 150mg QD, and 300mg QD) were combined as prespecified in SAP.
Groups:
- Phase 1: FT-2102 (Single Agent): Participants with AML or MDS received single agent FT-2102 orally BID in 28-day cycles at dose levels of 150 mg until MTD or MED achieved.
- Phase 1: Overall: Participants with AML or MDS received single agent (FT-2102), combination therapy (FT-2102 + azacitidine, FT-2102+ LDAC) starting at 150 mg BID dose level until MTD or MED achieved or treatment discontinuation.
Arm/Group | Phase 1: FT-2102 (Single Agent) | Phase 1: Total FT-2102 (Single Agent) | Phase 1: FT-2102 + Azacitidine (Combination Therapy) | Phase 1: Total FT-2102; FT-2102 + Azacitidine (Combination Therapy) | Phase 1: Overall | Phase 2: Cohort 1; FT-2102 (Single Agent) | Phase 2: Cohort 2; FT-2102 (Single Agent) | Phase 2: Cohort 3; FT-2102 (Single Agent) | Phase 2: Cohort 4; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 5; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 6; FT-2102 + Azacitidine (Combination Therapy) | Phase 2: Cohort 7; FT-2102 (Single Agent) | Phase 2: Cohort 8; FT-2102 + Azacitidine (Combination Therapy)
All-Cause Mortality (participants affected / at risk) | 4/16 | 11/31 | 9/39 | 10/46 | 21/78 | 50/153 | 0/18 | 2/5 | 3/20 | 6/21 | 7/20 | 4/10 | 2/11
Serious Adverse Events (participants affected / at risk) | 10/16 | 23/31 | 30/39 | 36/46 | 60/78 | 115/153 | 6/18 | 4/5 | 12/20 | 18/21 | 13/20 | 8/10 | 9/11
Other Adverse Events (participants affected / at risk) | 15/16 | 29/31 | 39/39 | 46/46 | 76/78 | 152/153 | 18/18 | 5/5 | 18/20 | 20/21 | 19/20 | 10/10 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: FT-2102 (Single Agent) (N=16) | Phase 1: Total FT-2102 (Single Agent) (N=31) | Phase 1: FT-2102 + Azacitidine (Combination Therapy) (N=39) | Phase 1: Total FT-2102; FT-2102 + Azacitidine (Combination Therapy) (N=46) | Phase 1: Overall (N=78) | Phase 2: Cohort 1; FT-2102 (Single Agent) (N=153) | Phase 2: Cohort 2; FT-2102 (Single Agent) (N=18) | Phase 2: Cohort 3; FT-2102 (Single Agent) (N=5) | Phase 2: Cohort 4; FT-2102 + Azacitidine (Combination Therapy) (N=20) | Phase 2: Cohort 5; FT-2102 + Azacitidine (Combination Therapy) (N=21) | Phase 2: Cohort 6; FT-2102 + Azacitidine (Combination Therapy) (N=20) | Phase 2: Cohort 7; FT-2102 (Single Agent) (N=10) | Phase 2: Cohort 8; FT-2102 + Azacitidine (Combination Therapy) (N=11)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute promyelocytic leukaemia differentiation syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2) | 4 (4) | 6 (6) | 14 (16) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Acute psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arterial stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspergillus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (2) | 1 (2) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial prostatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary tract disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catatonia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (3) | 2 (3) | 3 (4) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis microscopic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 3 (3) | 4 (4) | 5 (5) | 8 (8) | 25 (25) | 0 (0) | 1 (1) | 3 (3) | 4 (4) | 3 (3) | 1 (1) | 3 (3)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Familial mediterranean fever (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 6 (7) | 8 (12) | 10 (15) | 16 (22) | 23 (28) | 1 (1) | 2 (3) | 2 (4) | 4 (8) | 2 (2) | 2 (2) | 2 (2)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder perforation (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal angiectasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Human bocavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Klebsiella infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Labyrinthitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucormycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 7 (10) | 5 (6) | 7 (8) | 14 (18) | 14 (14) | 0 (0) | 1 (2) | 1 (1) | 4 (5) | 2 (2) | 1 (1) | 0 (0)
Pneumonia fungal (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia legionella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary mycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 3 (4) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Rectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Red blood cell count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 2 (3) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Septic shock (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Social stay hospitalisation (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 1 (2) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 2 (2) | 5 (6) | 3 (3) | 5 (5) | 10 (11) | 6 (6) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: FT-2102 (Single Agent) (N=16) | Phase 1: Total FT-2102 (Single Agent) (N=31) | Phase 1: FT-2102 + Azacitidine (Combination Therapy) (N=39) | Phase 1: Total FT-2102; FT-2102 + Azacitidine (Combination Therapy) (N=46) | Phase 1: Overall (N=78) | Phase 2: Cohort 1; FT-2102 (Single Agent) (N=153) | Phase 2: Cohort 2; FT-2102 (Single Agent) (N=18) | Phase 2: Cohort 3; FT-2102 (Single Agent) (N=5) | Phase 2: Cohort 4; FT-2102 + Azacitidine (Combination Therapy) (N=20) | Phase 2: Cohort 5; FT-2102 + Azacitidine (Combination Therapy) (N=21) | Phase 2: Cohort 6; FT-2102 + Azacitidine (Combination Therapy) (N=20) | Phase 2: Cohort 7; FT-2102 (Single Agent) (N=10) | Phase 2: Cohort 8; FT-2102 + Azacitidine (Combination Therapy) (N=11)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 5 (5) | 3 (3) | 4 (5) | 9 (10) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 7 (9) | 9 (11) | 10 (12) | 15 (17) | 0 (0) | 2 (2) | 2 (3) | 1 (1) | 2 (2) | 2 (3) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 4 (4) | 7 (9) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 3 (3) | 2 (2) | 3 (3) | 6 (6) | 7 (15) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acute promyelocytic leukaemia differentiation syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 4 (5) | 4 (5) | 6 (7) | 11 (11) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (9) | 3 (9) | 6 (6) | 7 (7) | 11 (17) | 18 (38) | 2 (5) | 1 (1) | 0 (0) | 2 (3) | 2 (3) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Angina bullosa haemorrhagica (Gastrointestinal disorders) | 1 (2) | 2 (3) | 1 (1) | 1 (1) | 3 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) | 5 (5) | 6 (6) | 9 (9) | 7 (7) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (2) | 2 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (9) | 8 (14) | 8 (14) | 13 (23) | 10 (14) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (8) | 5 (9) | 5 (8) | 5 (8) | 11 (18) | 14 (27) | 2 (3) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Aspergillus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 10 (14) | 11 (15) | 12 (16) | 30 (49) | 2 (2) | 1 (3) | 2 (2) | 3 (13) | 3 (4) | 1 (2) | 4 (11)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 5 (5) | 5 (5) | 6 (6) | 5 (7) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (5) | 5 (10) | 5 (10) | 9 (15) | 21 (29) | 4 (4) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 2 (4)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (5) | 3 (6) | 5 (8) | 6 (9) | 10 (16) | 9 (19) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 4 (8) | 4 (8) | 2 (2) | 3 (3) | 8 (12) | 8 (10) | 0 (0) | 1 (3) | 0 (0) | 3 (13) | 1 (1) | 1 (1) | 1 (6)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 5 (6) | 6 (7) | 7 (8) | 14 (15) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 1 (1) | 2 (2) | 2 (9)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain natriuretic peptide increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Chest X-ray abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 6 (10) | 6 (10) | 7 (11) | 6 (6) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (3) | 3 (3) | 3 (3) | 5 (6) | 6 (7) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 7 (7) | 24 (35) | 27 (41) | 34 (48) | 41 (51) | 4 (4) | 0 (0) | 5 (9) | 7 (9) | 10 (11) | 2 (2) | 7 (21)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 4 (4) | 5 (5) | 9 (9) | 6 (8) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5) | 15 (16) | 18 (19) | 23 (24) | 25 (33) | 3 (3) | 1 (1) | 4 (5) | 4 (5) | 3 (3) | 4 (5) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 7 (7) | 8 (12) | 10 (14) | 17 (21) | 26 (39) | 1 (1) | 0 (0) | 4 (5) | 4 (5) | 5 (7) | 3 (5) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (6) | 4 (7) | 6 (9) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 4 (5) | 4 (5) | 4 (5) | 6 (8) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 7 (8) | 16 (21) | 21 (29) | 29 (38) | 31 (36) | 1 (2) | 1 (1) | 5 (11) | 7 (8) | 5 (5) | 2 (3) | 4 (8)
Dizziness (Nervous system disorders) | 3 (5) | 7 (10) | 11 (16) | 11 (16) | 18 (26) | 10 (11) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 2 (2) | 1 (2)
Dry eye (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 5 (5) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 5 (5) | 6 (6) | 7 (7) | 7 (7) | 0 (0) | 1 (1) | 2 (5) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (5) | 4 (5) | 6 (7) | 11 (11) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 4 (4) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 7 (8) | 12 (22) | 13 (23) | 20 (31) | 31 (50) | 2 (3) | 2 (2) | 2 (2) | 1 (1) | 3 (4) | 2 (3) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Early satiety (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 3 (4) | 3 (4) | 6 (7) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 3 (4) | 3 (4) | 3 (4) | 12 (18) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 5 (6) | 7 (8) | 7 (8) | 12 (14) | 17 (32) | 0 (0) | 1 (1) | 4 (4) | 4 (4) | 1 (1) | 1 (1) | 3 (8)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 3 (5) | 3 (5) | 5 (7) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Eye haemorrhage (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 3 (4) | 4 (7) | 5 (8) | 8 (12) | 14 (14) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 6 (9) | 13 (16) | 16 (25) | 19 (28) | 32 (44) | 35 (47) | 6 (8) | 2 (2) | 6 (6) | 6 (7) | 7 (11) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 5 (7) | 5 (7) | 6 (8) | 12 (13) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (3) | 2 (2) | 2 (2) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 11 (24) | 2 (7) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4) | 4 (4) | 5 (5) | 6 (6) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival hypertrophy (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 3 (3) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 4 (5) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Haematuria (Renal and urinary disorders) | 3 (3) | 4 (4) | 5 (5) | 5 (5) | 9 (9) | 5 (5) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 1 (2)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 6 (7) | 13 (20) | 15 (22) | 21 (29) | 20 (27) | 6 (6) | 0 (0) | 6 (9) | 3 (3) | 1 (1) | 3 (3) | 2 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 3 (3) | 3 (3) | 6 (6) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 5 (5) | 7 (9) | 9 (15) | 14 (20) | 17 (31) | 0 (0) | 0 (0) | 4 (6) | 1 (1) | 2 (4) | 2 (2) | 2 (3)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 3 (3) | 4 (4) | 8 (8) | 6 (9) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (4) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (3) | 5 (5) | 7 (7) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 3 (6) | 5 (8) | 8 (11) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 7 (8) | 13 (18) | 16 (21) | 23 (29) | 33 (56) | 1 (1) | 3 (8) | 6 (11) | 1 (1) | 4 (4) | 1 (1) | 4 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 5 (5) | 5 (5) | 8 (8) | 8 (9) | 0 (0) | 1 (2) | 1 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 5 (5) | 5 (5) | 8 (8) | 6 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 4 (4) | 6 (7) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 4 (5) | 5 (5) | 5 (5) | 9 (10) | 7 (8) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 4 (4) | 4 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 3 (4) | 3 (4) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 4 (4) | 6 (6) | 5 (6) | 7 (8) | 13 (14) | 12 (13) | 3 (3) | 0 (0) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 2 (6)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (2) | 1 (2) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Lipase increased (Investigations) | 1 (1) | 1 (1) | 4 (6) | 4 (6) | 5 (7) | 10 (20) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (2) | 3 (3) | 4 (5) | 5 (11) | 8 (14) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 4 (5) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (3) | 0 (0) | 1 (1) | 3 (4) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 4 (4) | 6 (6) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 5 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (5) | 4 (4) | 4 (4) | 7 (9) | 6 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (2) | 3 (3) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 3 (3) | 4 (4) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 3 (4) | 3 (4) | 5 (6) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (11) | 14 (23) | 26 (37) | 32 (43) | 47 (68) | 59 (78) | 5 (7) | 3 (4) | 11 (14) | 9 (14) | 8 (11) | 2 (6) | 8 (12)
Neutrophil count decreased (Investigations) | 0 (0) | 3 (5) | 12 (35) | 14 (41) | 18 (47) | 21 (65) | 4 (10) | 0 (0) | 6 (7) | 5 (16) | 5 (14) | 2 (6) | 3 (11)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 8 (10) | 10 (12) | 12 (14) | 23 (36) | 2 (2) | 0 (0) | 3 (3) | 4 (4) | 4 (5) | 5 (5) | 1 (3)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (6) | 7 (8) | 7 (8) | 5 (5) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (2) | 2 (3) | 3 (3) | 4 (4) | 6 (7) | 6 (9) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 8 (13) | 8 (13) | 12 (17) | 13 (18) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (4)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 5 (5) | 5 (5) | 5 (5) | 5 (6) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 7 (9) | 7 (9) | 9 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 3 (4) | 7 (8) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 4 (7) | 8 (16) | 18 (67) | 20 (81) | 28 (97) | 31 (152) | 3 (4) | 1 (1) | 6 (34) | 9 (38) | 4 (32) | 1 (7) | 3 (20)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 4 (4) | 5 (5) | 6 (6) | 8 (8) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (2) | 2 (3) | 5 (9) | 5 (9) | 7 (12) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (2) | 1 (2) | 2 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 7 (8) | 8 (9) | 12 (13) | 8 (10) | 2 (3) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (2) | 2 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (5) | 9 (12) | 9 (14) | 11 (16) | 20 (28) | 35 (53) | 0 (0) | 1 (1) | 5 (9) | 1 (2) | 2 (3) | 3 (5) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 4 (4) | 4 (4) | 12 (12) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (4) | 0 (0) | 2 (6)
Red blood cell count decreased (Investigations) | 4 (6) | 6 (10) | 8 (26) | 11 (29) | 17 (39) | 40 (123) | 3 (7) | 1 (1) | 7 (27) | 5 (22) | 5 (26) | 2 (5) | 1 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 5 (6) | 5 (6) | 8 (9) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 2 (3) | 7 (7) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3) | 3 (3) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 5 (5) | 7 (7) | 12 (16) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 3 (3) | 5 (6) | 3 (4) | 3 (4) | 8 (10) | 5 (6) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 7 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 4 (5) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 5 (5) | 5 (5) | 10 (10) | 2 (4) | 0 (0) | 2 (2) | 2 (4) | 0 (0) | 1 (1) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (4) | 3 (4) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 3 (4) | 3 (4) | 4 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (4) | 3 (4) | 4 (5) | 14 (20) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 8 (12) | 14 (20) | 17 (23) | 25 (35) | 27 (35) | 2 (4) | 0 (0) | 10 (15) | 6 (6) | 6 (7) | 2 (3) | 4 (11)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 4 (4) | 5 (5) | 5 (5) | 7 (9) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 5 (6) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 2 (2) | 6 (9) | 8 (13) | 10 (15) | 4 (13) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 2 (3) | 3 (4) | 8 (10) | 10 (12) | 13 (16) | 36 (56) | 1 (1) | 2 (6) | 3 (6) | 3 (3) | 4 (6) | 0 (0) | 1 (1)
Abdominal rigidity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Administration site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Affective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Aortic calcification (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Articular calcification (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Catheter site rash (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (2) | 5 (6) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronavirus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 3 (5) | 3 (5) | 4 (6) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endotheliomatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterobacter bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterococcus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophilic colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Essential tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flat affect (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Genital erythema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 2 (3) | 2 (3) | 2 (3) | 2 (3) | 4 (6) | 4 (9) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (11) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperferritinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypogammaglobulinaemia (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Klebsiella infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lower respiratory tract infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macular fibrosis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Motor dysfunction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 3 (3) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal dryness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 7 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 8 (11) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 4 (5) | 4 (5) | 4 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seronegative arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 2 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 4 (4) | 4 (4) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue dysplasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 4 (5) | 4 (5) | 5 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Visual field defect (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood blister (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related thrombosis (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 2 (4) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/74/NCT02719574/Prot_000.pdf
  • Statistical Analysis Plan (2015-04-13): https://cdn.clinicaltrials.gov/large-docs/74/NCT02719574/SAP_001.pdf